#### 1 TITLE PAGE



VERTEX PHARMACEUTICALS INCORPORATED

# **Clinical Study Protocol**

A Phase 3b, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-445/Tezacaftor/Ivacaftor in Cystic Fibrosis Subjects, Homozygous for *F508del* 

> Vertex Study Number: VX18-445-109 EudraCT Number: 2019-001735-31

**Date of Protocol:** 30 May 2019 (Version 1.0)

Vertex Pharmaceuticals Incorporated 50 Northern Avenue Boston, MA 02210-1862, USA

#### **CONFIDENTIAL**

This document contains confidential information. Any use, distribution, or disclosure without the prior written consent of Vertex Pharmaceuticals Incorporated is strictly prohibited except to the extent required under applicable laws or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them.

#### 2 PROTOCOL SYNOPSIS

**Title** A Phase 3b, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-445/Tezacaftor/Ivacaftor in Cystic Fibrosis Subjects, Homozygous

for F508del

**Brief Title** A Study Evaluating the Efficacy and Safety of VX-445/Tezacaftor/Ivacaftor in Cystic

Fibrosis Subjects, Homozygous for F508del

Clinical Phase and Clinical Study Type Phase 3b, efficacy and safety

#### **Objectives Primary Objective**

To evaluate the efficacy of VX-445/tezacaftor (TEZ)/ivacaftor (IVA) in cystic fibrosis (CF) subjects, homozygous for *F508del* (F/F).

#### **Secondary Objectives**

- To evaluate the safety of VX-445/TEZ/IVA
- To evaluate the pharmacodynamics (PD) of VX-445/TEZ/IVA

#### **Endpoints Primary Endpoint**

 Absolute change in CF Questionnaire-Revised (CFQ-R) respiratory domain score from baseline through Week 24

#### **Key Secondary Endpoint**

• Absolute change in percent predicted forced expiratory volume in 1 second (ppFEV<sub>1</sub>) from baseline through Week 24

#### **Secondary Endpoints**

- Absolute change in sweat chloride (SwCl) from baseline through Week 24
- Safety and tolerability assessments based on adverse events (AEs), clinical laboratory values, ECGs, vital signs, and pulse oximetry

**Number of Subjects** Up to approximately 158 subjects will be randomized (1:1) to either the VX-445/TEZ/IVA group or the TEZ/IVA group.

**Study Population** Male and female CF subjects who are 12 years of age or older and have an F/F genotype

Investigational Drug During the TEZ/IVA Run-in Period, study drug refers to TEZ/IVA and IVA.

During the Treatment Period, study drug refers to VX-445/TEZ/IVA and matching placebo, TEZ/IVA and matching placebo, and IVA.

Active study drugs will be orally administered as fixed-dose combination (FDC) film-coated tablets (either VX-445/TEZ/IVA or TEZ/IVA) in the morning and as a film-coated IVA tablet in the evening.

Active substance: VX-445/TEZ (VX-661)/IVA (VX-770)

Activity: CFTR corrector, CFTR corrector, and CFTR potentiator

**Strength:** 100 mg/50 mg/75 mg

**Active substance:** TEZ (VX-661)/ IVA (VX-770) **Activity:** CFTR corrector and CFTR potentiator

Strength: 100 mg/150 mg

Active substance: IVA (VX-770) Activity: CFTR potentiator

Strength: 150 mg

#### **Study Duration**

The total study duration is approximately 36 weeks (4 weeks for the Screening Period, 4 weeks for the TEZ/IVA Run-in Period, 24 weeks for the Treatment Period, and 4 weeks for the Safety Follow-up Period).

#### **Study Design**

This is a Phase 3b, randomized, double-blind, active-controlled, parallel-group, multicenter study (Figure 2-1).

Figure 2-1 Schematic of the Study Design



IVA: ivacaftor; N: number of subjects; TEZ: tezacaftor

Note: The Safety Follow-up Visit is not required for subjects who complete the Week 24 Visit and have enrolled in an open-label study within 28 days after the last dose of study drug.

In the TEZ/IVA Run-in Period, all subjects will receive TEZ 100 mg once daily (qd)/IVA 150 mg every 12 hours (q12h). After completing the TEZ/IVA Run-in Period, subjects will be randomized (1:1) to the VX-445/TEZ/IVA group or TEZ/IVA group for the Treatment Period (Table 2-1).

Table 2-1 Treatment Period Groups and Dosages

| <b>Treatment Group</b> | VX-445 Dosage | TEZ Dosage | IVA Dosage |
|------------------------|---------------|------------|-------------|
| VX-445/TEZ/IVA | 200 mg qd | 100 mg qd | 150 mg q12h |
| TEZ/IVA | 0 mg qd | 100 mg qd | 150 mg q12h |

IVA: ivacaftor; q12h: every 12 hours; qd: once daily; TEZ: tezacaftor Randomization will be stratified by ppFEV<sub>1</sub> determined during the TEZ/IVA Run-in Period (Day -14 assessment; <70 versus  $\geq$ 70), age at the Screening Visit (<18 versus  $\geq$ 18 years of age), and whether the subject is receiving CFTR modulator treatment at the Screening Visit (yes versus no). If the Day -14 ppFEV<sub>1</sub> value is not valid or not

available, the most recent available ppFEV<sub>1</sub> value will be used for stratification.

**Assessments** Efficacy: CFQ-R, spirometry

PD: SwCl

**Safety:** AEs, clinical laboratory assessments, ECGs, vital signs, pulse oximetry, ophthalmologic examinations, and physical examinations

#### Statistical Analyses Statistical Methods/Analyses

The baseline value, unless otherwise specified, will be defined as the most recent non-missing measurement collected before the first dose of study drug in the Treatment Period (i.e., the Day 1 Visit). The TEZ/IVA Run-in Period is intended to establish a reliable on-treatment (TEZ/IVA) baseline for comparison during the Treatment Period.

The primary efficacy endpoint is the absolute change in CFQ-R respiratory domain score from baseline through Week 24. The primary null hypothesis to be tested is that the mean absolute change in CFQ-R respiratory domain score from baseline through Week 24 is the same for the VX-445/TEZ/IVA and TEZ/IVA groups. The null hypothesis will be tested at a 2-sided significance level of 0.05.

Assuming a within-group SD of 18 and a treatment difference of 10 between VX-445/TEZ/IVA and TEZ/IVA, a sample size of 71 subjects completing the Treatment Period in each group for a total of 142 subjects will have approximately 90% power for the CFQ-R respiratory domain score hypothesis testing, based on a 2-sample t-test at a significance level of 0.05. Assuming a 10% dropout rate, up to approximately 158 subjects will be enrolled.

The primary analysis for CFQ-R will be based on a mixed-effects model for repeated measures (MMRM). The primary result obtained from the model will be the estimated treatment difference through Week 24. The treatment difference at each post-baseline visit, obtained from the model, will also be provided.

A hierarchical fixed-sequence testing procedure will be used to control the overall family-wise type I error for the testing of the primary endpoint and key secondary endpoint.

The safety endpoints include AEs, clinical laboratory values, ECGs, vital signs, and pulse oximetry through the Safety Follow-up Visit. The safety analysis will be descriptive only.

### 3 SCHEDULE OF ASSESSMENTS

Schedules of assessments are in Table 3-1 and Table 3-2.

All visits are to be scheduled relative to the Day 1 Visit (first dose of randomized study drug in the Treatment Period). For example, the Week 4 ( $\pm$  5 days) Visit would occur after 4 weeks of study drug administration in the Treatment Period has been completed.

The Cystic Fibrosis Questionnaire—Revised (CFQ-R) must be completed before any other assessment (except signing of ICF) at relevant clinic visits. Remaining assessments may be performed in any order when more than 1 assessment is required at a particular time point. All assessments will be performed before study drug dosing (Section 9.6.1), unless noted otherwise.

Table 3-1 Study VX18-445-109: Screening

| Event/Assessment | Screening Visit<br>Day -56 to Day -29 | Comments |
|---|---|---|
| ICF and assent (when applicable) | X | |
| Inclusion and exclusion criteria review | X | |
| Demographics | X | |
| Medical history | X | |
| CFQ-R | X | Completed before the start of any other assessments (except signing ICF) scheduled for that visit. |
| CFTR genotype | X | If the screening CFTR genotype result is not received before enrollment, a previous <i>CFTR</i> genotype laboratory report may be used to establish eligibility. Subjects who have been enrolled and whose screening genotype does not confirm eligibility must be discontinued from the study. |
| FSH | X | Measured for any suspected postmenopausal female with at least 12 months of continuous spontaneous amenorrhea. |
| Serum pregnancy test (all female subjects) | X | |
| Hematology | X | |
| Coagulation | X | |
| Serum chemistry | X | |
| Urinalysis | X | |
| Weight and height | X | Measured with shoes off. |
| Ophthalmologic examination | X | Only conducted for subjects who are <18 years of age on the date of informed consent. |
| Complete physical examination | X | |
| Vital signs and pulse oximetry | X | Collected after the subject has been at rest for at least 5 minutes. |
| Standard 12-lead ECG | X | Performed after the subject has been at rest for at least 5 minutes. |
| Spirometry | X | Performed pre- or post-bronchodilator. |
| Medications review | X | |
| Sweat chloride | X | |
| AEs and SAEs | Continuous from signing<br>of ICF through Safety<br>Follow-up Visit | |

AE: adverse event; CFQ-R: Cystic Fibrosis Questionnaire-Revised; FSH: follicle stimulating hormone; ICF: informed consent form; SAE: serious adverse event

Page 7 of 60 Protocol VX18-445-109, Version 1.0

| | | A Run-in<br>4 weeks) | | , | Т | reatment Po | eriod (24 we | eks) | | | | Safety<br>Follow-up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Event/<br>Assessment <sup>a</sup> | Day -28<br>± 1 day | Day -14<br>(Day -15<br>to<br>Day -3) | Day 1 <sup>d</sup> | Day 15 ± 3 days | Week 4<br>± 5 days | Week 8<br>± 5 days | Week 12<br>± 5 days | Week 16<br>± 5 days | Week 20<br>± 5 days | Week 24<br>± 5 days | ETT<br>Visit <sup>b</sup> | Visit <sup>c</sup> (28 ± 7 Days After Last Dose of Study Drug) | Comments |
| Clinic visit | X | X | X | X | X | X | | X | | X | X | X | |
| Telephone contact | | | | | | | X | | X | | | | Assess the subject's status, any AEs, concomitant medications, treatments, and procedures. |
| Inclusion and exclusion criteria confirmation | X | | | | | | | | | | | | |
| CFQ-R | | | X | | X | X | | X | | Х | X | X | Completed before any other assessments scheduled at relevant visits (Section 11.4.1). |
| Weight and height | X | | X | X | X | X | | X | | X | X | X | Measured with shoes off. |

X

X

X

X

Height will only be collected for subjects ≤21 years of age on the date of informed consent (Section 11.4.3).

Subjects <18 years of age on

the date of informed consent and who completed at least 12 weeks of study drug treatment will have a single ophthalmologic examination at either the ETT or Week 24 Visit, whichever comes first

Symptom directed physical

examinations may be

performed at any time if deemed necessary by the investigator (Section 11.5.3).

(Section 11.5.6).

X

X

X

Ophthalmologic

Complete physical

examination

examination

All assessments will be performed before dosing unless noted otherwise.

If a subject prematurely discontinues study drug treatment, an ETT Visit should be scheduled as soon as possible after the decision to discontinue treatment. Subjects who prematurely discontinue treatment during the Treatment Period will continue to complete all scheduled study visits for assessments following completion of the ETT Visit.

The Safety Follow-up Visit is required for all subjects, unless the subject completes the Week 24 Visit and has enrolled in a separate open-label study within 28 days after the last dose of study drug. If an ETT Visit occurs 3 weeks or later following the last dose of study drug, then the ETT Visit replaces the Safety Follow-up Visit.

To enter the Treatment Period, conditions for entry must be satisfied.

Protocol VX18-445-109, Version 1.0

| Table 3-2 | Study VX18-445-109: Treatment Period and Safety Follow-up Visit |
|-----------|-----------------------------------------------------------------|
|-----------|-----------------------------------------------------------------|

| 1 able 3-2 | Study VX | | 09. ITE | atiliciit f | criou all | u Saiety | i onow-u | h visit | | | 1 | G.C. | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | A Run-in<br>4 weeks) | | | Т | reatment P | eriod (24 we | eks) | | | | Safety<br>Follow-up | |
| Event/<br>Assessment <sup>a</sup> | Day -28<br>± 1 day | Day -14<br>(Day -15<br>to<br>Day -3) | Day 1 <sup>d</sup> | Day 15 ± 3 days | Week 4<br>± 5 days | Week 8<br>± 5 days | Week 12<br>± 5 days | Week 16<br>± 5 days | Week 20<br>± 5 days | Week 24<br>± 5 days | ETT<br>Visit <sup>b</sup> | Visit <sup>c</sup> (28 ± 7 Days After Last Dose of Study Drug) | Comments |
| Pregnancy testing<br>(all female<br>subjects) | urine | | urine | urine | urine | urine | urine | urine | urine | urine | serum | serum | At telephone contacts, a urine pregnancy test will be performed with a home kit provided by the study site. Results will be reported to the site by telephone. |
| Standard 12-lead<br>ECG | X | | X | | | X | | | | X | X | X | Performed after subject has been at rest for at least 5 minutes (Section 11.5.5). |
| Vital signs and pulse oximetry | X | | X | X | X | X | | X | | X | X | X | Performed after subject has been at rest for at least 5 minutes (Sections 11.5.3 and 11.5.4). |
| Spirometry | | X | X | X | X | X | | X | | X | X | X | Should be performed pre-bronchodilator and at approximately the same time at each visit (Section 11.4.2). |
| Sweat chloride | | X | X | | X | X | | | | X | X | | At each time point, 2 samples will be collected (1 from each arm, Section 11.3). |
| Urinalysis | X | | X | | | | | | | X | X | | |
| Hematology | X | | X | X | X | X | | X | | X | X | X | |
| Coagulation | X | | X | | | | | | | X | X | X | |
| Serum chemistry | X | | X | X | X | X | | X | | X | X | X | |
| Run-in TEZ/IVA<br>dosing | on D | to evening<br>Pay -1 | | | | | | | | | | | |
| Run-in TEZ/IVA<br>drug count | X | X | X | | | | | | | | | | |
| Randomization | | | X | | | | | | | | | | May occur on Day -1 or Day 1 after eligibility for entry into the Treatment Period has been satisfied. |
| Randomized study drug dosing | | | | | ay 1 through | evening before | ore Week 24 | | | | | | |
| Randomized study drug count | 4:1- I | | X | X | X | X | | X | | X | X | | |

Vertex Pharmaceuticals Incorporated

Protocol VX18-445-109, Version 1.0 Page 9 of 60

| | TEZ/IVA Run-in Period (4 weeks) Treatment Period (24 weeks) Safety Follow-up | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Event/<br>Assessment <sup>a</sup> | Day -28<br>± 1 day | Day -14<br>(Day -15<br>to<br>Day -3) | Day 1 <sup>d</sup> | Day 15<br>± 3 days | Week 4<br>± 5 days | Week 8<br>± 5 days | Week 12<br>± 5 days | Week 16<br>± 5 days | Week 20<br>± 5 days | Week 24<br>± 5 days | ETT<br>Visit <sup>b</sup> | Visit <sup>c</sup> (28 ± 7 Days After Last Dose of Study Drug) | Comments |
| Medications<br>review | | Continuous from signing of ICF through completion of study participation Completion of study participation participation is defined in Section 9.1.7. | | | | | | | | | | | |
| Treatment and procedures review | | Continuous from signing of ICF through completion of study participation | | | | | | | | | Completion of study participation is defined in Section 9.1.7. | | |
| AEs and SAEs | | Continuous from signing of ICF through completion of study participation | | | | | | | | Completion of study participation is defined in Section 9.1.7. | | | |

# 4 TABLE OF CONTENTS

| 1 | The rage | |
|---|------------------------------------------------------|------|
| 2 | Protocol Synopsis | |
| 3 | Schedule of Assessments | 5 |
| 4 | Table of Contents | |
| | List of Tables. | . 13 |
| | List of Figures | |
| | List of Abbreviations | . 14 |
| 5 | Introduction | . 16 |
| | 5.1 Background | . 16 |
| | 5.2 Rationale for the Present Study | . 16 |
| 6 | Study Objectives | . 17 |
| | 6.1 Primary Objective | . 17 |
| | 6.2 Secondary Objectives | . 17 |
| 7 | Study Endpoints | . 17 |
| | 7.1 Primary Endpoint | . 17 |
| | 7.2 Key Secondary Endpoint | . 17 |
| | 7.3 Secondary Endpoints | . 17 |
| 8 | Study Population | . 17 |
| | 8.1 Inclusion Criteria | . 17 |
| | 8.2 Exclusion Criteria | . 18 |
| 9 | Study Implementation | . 19 |
| | 9.1 Study Design | . 19 |
| | 9.1.1 Screening | |
| | 9.1.1.1 Repetition of Screening Assessment(s) | . 21 |
| | 9.1.1.2 Rescreening | |
| | 9.1.1.3 Extension of Screening Period Window | . 21 |
| | 9.1.2 Tezacaftor/Ivacaftor Run-in Period | . 21 |
| | 9.1.3 Treatment Period | |
| | 9.1.4 Follow-up | |
| | 9.1.5 Early Termination of Treatment | |
| | 9.1.5.1 Discontinuation During the Run-in Period | |
| | 9.1.5.2 Discontinuation During the Treatment Period | |
| | 9.1.6 Lost to Follow-up | |
| | 9.1.7 Completion of Study Participation | |
| | 9.2 Method of Assigning Subjects to Treatment Groups | . 23 |
| | 9.3 Rationale for Study Elements | . 24 |
| | 9.3.1 Study Design | |
| | 9.3.2 Study Population. | |
| | 9.3.3 Study Drug Dose | |
| | 9.3.4 Rationale for Study Assessments | . 24 |
| | 9.4 Study Restrictions | |
| | 9.4.1 Prohibited Medications | |
| | 9.5 Prior and Concomitant Medications | . 25 |
| | 9.6 Administration | . 26 |

| 9.6.1 Dosing | |
|--------------------------------------------|-----------------|
| 9.6.2 Missed Doses | 27 |
| 9.7 Dose Modification for Toxicity | 27 |
| 9.8 Study Drug Interruption and Stopping | g Rules |
| | 27 |
| 9.8.2 Rash | 28 |
| 9.9 Removal of Subjects | |
| 9.10 Replacement of Subjects | |
| 10 Study Drug Information and Managem | ent29 |
| 10.2 Packaging and Labeling | |
| 10.3 Study Drug Supply, Storage, and Har | ndling30 |
| | 30 |
| 10.5 Disposal, Return, or Retention of Uni | used Drug31 |
| 10.6 Compliance | 31 |
| 10.7 Blinding and Unblinding | 31 |
| 10.7.1 Blinding | 31 |
| 10.7.2 Unblinding | |
| 11 Assessments | 33 |
| 11.1 Timing of Assessments | |
| 11.2 Subject and Disease Characteristics | |
| 11.3 Pharmacodynamics: Sweat Chloride. | |
| 11.4.1 Cystic Fibrosis Questionnaire-R | evised |
| 11.4.2 Spirometry | |
| 11.5 Safety | |
| 11.5.1 Adverse Events | |
| 11.5.2 Clinical Laboratory Assessment | s |
| | Signs |
| 11.5.4 Pulse Oximetry | |
| 11.5.5 Electrocardiograms | |
| 11.5.7 Contraception and Pregnancy | |
| • | |
| 11.5.7.2 Pregnancy | 40 |
| 12 Statistical and Analytical Plans | 40 |
| <u> </u> | 40 |
| • | 41 |
| | 41 |
| | 41 |
| $oldsymbol{arepsilon}$ | 42 |
| | Characteristics |
| | ications |
| 12.3.2.4 Study Drug Exposure and C | ompliance 43 |

| 12.3.3 Efficacy and Pharmacodynamic Analyses 4 12.3.3.1 Analysis of Primary Endpoint 4 12.3.3.2 Analysis of Key Secondary Endpoint 4 12.3.3.3 Analysis of Secondary Endpoint 4 12.3.3.4 Multiplicity Adjustment 4 12.3.4 Safety Analysis 4 12.3.4.1 Adverse Events 4 12.3.4.2 Clinical Laboratory Assessments 4 12.3.4.2 Clinical Laboratory Assessments 4 12.3.4.3 Electrocardiogram 4 12.3.4.5 Pulse Oximetry 4 12.3.4.6 Physical Examination 4 12.3.4.5 Pulse Oximetry 4 12.3.4.6 Physical Examination 4 12.3.5.1 Interim Analysis 4 12.3.5.2 IDMC Analysis 4 12.3.5.2 IDMC Analysis 4 13.1.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting 4 13.1.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting 4 13.1.1.1 Definition of an Adverse Event 4 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2 Experiting and Documentation of Serious Adverse Events 5 13.1.2 Experiting and Investigator Safety Letters 5 13.2.2 Experiting and Investigator Safety Letters 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Experiting and Investigator Safety Letters 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.2.5 Electronic Data Capture 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | | Important Protocol Deviations | |
|---|---|---|---|---|
| 12.3.3.1 Analysis of Frimary Endpoint | | 12.3.3 Eff | ficacy and Pharmacodynamic Analyses | 43 |
| 12.3.3.3 Analysis of Secondary Endpoint 4 12.3.4 Safety Analysis 4 12.3.4 Safety Analysis 4 12.3.4.1 Adverse Events | | | | |
| 12.3.4 Multiplicity Adjustment 4 12.3.4.1 Adverse Events. 4 12.3.4.2 Clinical Laboratory Assessments. 4 12.3.4.3 Electrocardiogram 4 12.3.4.5 Pulse Oximetry. 4 12.3.4.5 Pulse Oximetry. 4 12.3.4.6 Physical Examination. 4 12.3.5.1 Interim and IDMC Analyses. 4 12.3.5.2 IDMC Analysis. 4 13.1.2.3.5.2 IDMC Analysis. 4 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting. 4 13.1.1 Adverse Events 4 13.1.1.1 Definition of an Adverse Event. 4 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Causality 4 13.1.1.5 Adverse Event Causality 4 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2 | | 12.3.3.2 | Analysis of Key Secondary Endpoint | 44 |
| 12.3.4 Safety Analysis 4 12.3.4.2 Clinical Laboratory Assessments 4 12.3.4.3 Electrocardiogram 4 12.3.4.4 Vital Signs 4 12.3.4.5 Pulse Oximetry 4 12.3.4.6 Physical Examination 4 12.3.5 Interim and IDMC Analyses 4 12.3.5.1 Interim Analysis 4 12.3.5.2 IDMC Analysis 4 12.3.5.1 Interim Analysis 4 13.1.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting 4 13.1.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting 4 13.1.1.1 Definition of an Adverse Event 4 13.1.1.1 Definition of an Adverse Event 4 13.1.1.1 Adverse Event Severity 4 13.1.1.1 Adverse Event Severity 4 13.1.1.1 Adverse Event Causality 4 13.1.1.2 Strious Adverse Event 5 13.1.1.3 Treatment Given 5 13.1.1 Adverse Event Severity 4 13.1.1.2 Serious Adverse Event 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2.4 Administrative Requirements 5 13.2.5 Subject Information and Informed Consent 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.2.9 End of Study 5 13.20 Subject Privacy 5 13.21 Ectrical Consideration 5 13.22 Subject Information 5 13.23 Data Quality Assurance 5 13.44 Monitoring 5 13.55 Electronic Data Capture 5 13.65 Confidentiality and Disclosure 5 13.66 Confidentiality and Disclosure 5 13.67 Confidentiality and Disclosure 5 13.68 Confidentiality and Disclosure 5 13.60 C | | 12.3.3.3 | Analysis of Secondary Endpoint | 44 |
| 12.3.4.1 Adverse Events | | 12.3.3.4 | Multiplicity Adjustment | 44 |
| 12.3.4.2 Clinical Laboratory Assessments 4 12.3.4.3 Electrocardiogram 4 12.3.4.4 Vital Signs 4 12.3.4.5 Pulse Oximetry 4 12.3.5.1 Interim and IDMC Analyses 4 12.3.5.2 Interim Analysis 4 12.3.5.2 IDMC Analysis 4 13 Procedural, Ethical, Regulatory, and Administrative Considerations 4 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting 4 13.1.1 Definition of an Adverse Event 4 13.1.1.1 Definition of an Adverse Event 4 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.2.2 Subject Information and Informed Consent 5 13.2.1 Ethic | | 12.3.4 Sa | fety Analysis | 45 |
| 12.3.4.3 Electrocardiogram | | 12.3.4.1 | Adverse Events | 45 |
| 12.3.4.4 Vital Signs 4 12.3.4.5 Pulse Oximetry 4 12.3.5 Interim and IDMC Analyses 4 12.3.5.1 Interim Analysis 4 12.3.5.2 IDMC Analysis 4 13 Procedural, Ethical, Regulatory, and Administrative Considerations 4 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting 4 13.1.1 Adverse Events 4 13.1.1.1 Definition of an Adverse Event 4 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 | | 12.3.4.2 | Clinical Laboratory Assessments | 46 |
| 12.3.4.5 Pulse Oximetry. 4 12.3.4.6 Physical Examination. 4 12.3.5.1 Interim and IDMC Analysis. 4 12.3.5.2 IDMC Analysis. 4 13.1 Procedural, Ethical, Regulatory, and Administrative Considerations. 4 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting. 4 13.1.1 Definition of an Adverse Event. 4 13.1.1.1 Definition of an Adverse Event. 4 13.1.1.2 Clinically Significant Assessments. 4 13.1.1.3 Documentation of Adverse Events. 4 13.1.1.4 Adverse Event Severity. 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2 Serious Adverse Events 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.2.2 Reporting and Investigator Safety Letters 5 <t< th=""><td></td><td>12.3.4.3</td><td>Electrocardiogram</td><td> 46</td></t<> | | 12.3.4.3 | Electrocardiogram | 46 |
| 12.3.4.6 Physical Examination 4 12.3.5 Interim and IDMC Analyses 4 12.3.5.1 Interim Analysis 4 12.3.5.2 IDMC Analysis 4 13 Procedural, Ethical, Regulatory, and Administrative Considerations 4 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting 4 13.1.1 Adverse Events 4 13.1.1.1 Definition of an Adverse Event 4 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.8 End of Study< | | 12.3.4.4 | Vital Signs | 47 |
| 12.3.5 Interim and IDMC Analyses 4 12.3.5.1 Interim Analysis 4 13 Procedural, Ethical, Regulatory, and Administrative Considerations 4 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting 4 13.1.1 Adverse Events 4 13.1.1.1 Definition of an Adverse Event 4 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance | | 12.3.4.5 | Pulse Oximetry | 47 |
| 12.3.5.1 Interim Analysis 4 12.3.5.2 IDMC Analysis 4 13 Procedural, Ethical, Regulatory, and Administrative Considerations 4 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting 4 13.1.1 Adverse Events 4 13.1.1.1 Definition of an Adverse Event 4 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.2.2 Expedited Reporting and Investigator Safety Letters 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent | | 12.3.4.6 | Physical Examination | 47 |
| 12.3.5.2 IDMC Analysis 4 13 Procedural, Ethical, Regulatory, and Administrative Considerations 4 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting 4 13.1.1 Adverse Events 4 13.1.1.1 Definition of an Adverse Event 4 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2 Serious Adverse Events 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2 Administrative Requirements 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.7 Study Termination 5 13.2.8 End of | | 12.3.5 Int | erim and IDMC Analyses | 47 |
| 13 Procedural, Ethical, Regulatory, and Administrative Considerations 4 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting 4 13.1.1 Adverse Events 4 13.1.1.1 Definition of an Adverse Event 4 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2 Administrative Requirements 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assuran | | 12.3.5.1 | Interim Analysis | 47 |
| 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting 4 13.1.1 Adverse Events 4 13.1.1.1 Definition of an Adverse Event 4 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2 Serious Adverse Events 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2 Administrative Requirements 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 < | | | | |
| Reporting 4 13.1.1 Adverse Events 4 13.1.1.1 Definition of an Adverse Event 4 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.2.1 Treatment Given 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 <td>13</td> <td>Procedural,</td> <td>, Ethical, Regulatory, and Administrative Considerations</td> <td> 48</td> | 13 | Procedural, | , Ethical, Regulatory, and Administrative Considerations | 48 |
| 13.1.1 Adverse Events 4 13.1.1.1 Definition of an Adverse Event 4 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2 Serious Adverse Events 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | | | |
| 13.1.1.1 Definition of an Adverse Event. 4 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events. 4 13.1.1.4 Adverse Event Severity. 4 13.1.1.5 Adverse Event Causality. 4 13.1.1.6 Study Drug Action Taken. 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given. 5 13.1.2 Serious Adverse Events. 5 13.1.2.1 Definition of a Serious Adverse Event. 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 <td></td> <td>-</td> <td></td> <td></td> | | - | | |
| 13.1.1.2 Clinically Significant Assessments 4 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2 Serious Adverse Events 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 | | _ | | _ |
| 13.1.1.3 Documentation of Adverse Events 4 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2 Serious Adverse Events 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2.1 Ethical Considerations 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.8 End of Study 5 13.2.8 End of Study 5 13.5 Electronic Data Capture 5 13.6 <td< th=""><td></td><td>13.1.1.1</td><td></td><td></td></td<> | | 13.1.1.1 | | |
| 13.1.1.4 Adverse Event Severity 4 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2 Serious Adverse Events 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2 Administrative Requirements 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | 13.1.1.2 | | |
| 13.1.1.5 Adverse Event Causality 4 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2 Serious Adverse Events 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | 13.1.1.3 | | |
| 13.1.1.6 Study Drug Action Taken 5 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2 Serious Adverse Events 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2 Administrative Requirements 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | | | |
| 13.1.1.7 Adverse Event Outcome 5 13.1.1.8 Treatment Given 5 13.1.2 Serious Adverse Events 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2 Administrative Requirements 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | | · | |
| 13.1.1.8 Treatment Given. 5 13.1.2 Serious Adverse Events. 5 13.1.2.1 Definition of a Serious Adverse Event. 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events. 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters. 5 13.2 Administrative Requirements. 5 13.2.1 Ethical Considerations. 5 13.2.2 Subject Information and Informed Consent. 5 13.2.3 Investigator Compliance. 5 13.2.4 Access to Records. 5 13.2.5 Subject Privacy. 5 13.2.6 Record Retention. 5 13.2.7 Study Termination. 5 13.2.8 End of Study. 5 13.3 Data Quality Assurance. 5 13.4 Monitoring. 5 13.5 Electronic Data Capture. 5 13.6 Confidentiality and Disclosure. 5 | | | • | |
| 13.1.2 Serious Adverse Events 5 13.1.2.1 Definition of a Serious Adverse Event 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2 Administrative Requirements 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | | | |
| 13.1.2.1 Definition of a Serious Adverse Event. 5 13.1.2.2 Reporting and Documentation of Serious Adverse Events. 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters. 5 13.2 Administrative Requirements. 5 13.2.1 Ethical Considerations. 5 13.2.2 Subject Information and Informed Consent. 5 13.2.3 Investigator Compliance. 5 13.2.4 Access to Records. 5 13.2.5 Subject Privacy. 5 13.2.6 Record Retention. 5 13.2.7 Study Termination. 5 13.2.8 End of Study. 5 13.3 Data Quality Assurance. 5 13.4 Monitoring. 5 13.5 Electronic Data Capture. 5 13.6 Confidentiality and Disclosure. 5 | | | | |
| 13.1.2.2 Reporting and Documentation of Serious Adverse Events 5 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2 Administrative Requirements 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | | | |
| 13.1.2.3 Expedited Reporting and Investigator Safety Letters 5 13.2 Administrative Requirements 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | | | |
| 13.2 Administrative Requirements 5 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | | | |
| 13.2.1 Ethical Considerations 5 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | | | |
| 13.2.2 Subject Information and Informed Consent 5 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | _ | 1 | |
| 13.2.3 Investigator Compliance 5 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | | | |
| 13.2.4 Access to Records 5 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | | | |
| 13.2.5 Subject Privacy 5 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | | | |
| 13.2.6 Record Retention 5 13.2.7 Study Termination 5 13.2.8 End of Study 5 13.3 Data Quality Assurance 5 13.4 Monitoring 5 13.5 Electronic Data Capture 5 13.6 Confidentiality and Disclosure 5 | | | | |
| 13.2.7 Study Termination513.2.8 End of Study513.3 Data Quality Assurance513.4 Monitoring513.5 Electronic Data Capture513.6 Confidentiality and Disclosure5 | | | | |
| 13.2.8 End of Study513.3 Data Quality Assurance513.4 Monitoring513.5 Electronic Data Capture513.6 Confidentiality and Disclosure5 | | | | |
| 13.3 Data Quality Assurance513.4 Monitoring513.5 Electronic Data Capture513.6 Confidentiality and Disclosure5 | | | | |
| 13.4 Monitoring513.5 Electronic Data Capture513.6 Confidentiality and Disclosure5 | | | | |
| 13.5 Electronic Data Capture513.6 Confidentiality and Disclosure5 | | | | |
| 13.6 Confidentiality and Disclosure | | | · · | |
| | | | <u> </u> | |
| 13.7 Publications and Clinical Study Report | | 13.7 Publicat | tions and Clinical Study Report | 55 |

| 13.7.1 | Publication of Study Results | 55 |
|---|---|---|
| | Clinical Study Report | |
| | ices | |
| | l Signature Pages | |
| | onsor Signature Page | |
| - | estigator Signature Page | |
| List of Tab | les | |
| Table 2-1 | Treatment Period Groups and Dosages | 3 |
| Table 3-1 | Study VX18-445-109: Screening | |
| Table 3-2 | Study VX18-445-109: Treatment Period and Safety Follow-up Visit | |
| Table 9-1 | Treatment Period Groups and Dosages | |
| Table 9-2 | Prohibited Medications | |
| Table 10-1 | Study Drug: Strength/Dosing Form/Route | |
| Table 11-1 | Safety Laboratory Test Panels | |
| Table 11-2 | Acceptable Methods of Contraception | |
| Table 13-1 | Grading of AE Severity | |
| Table 13-2 | Classifications for AE Causality | |
| Table 13-3 | Classifications for Study Drug Action Taken With Regard to an AE | |
| Table 13-4 | Classifications for Outcome of an AE | |
| List of Fig | ures | |
| Figure 2-1 | Schematic of the Study Design | 3 |
| Figure 9-1 | Schematic of the Study Design | 20 |

# **List of Abbreviations**

| AE adverse event ALP alkaline phosphatase ALT alamine transaminase AST aspartate transaminase AST aspartate transaminase CF eystic fibrosis CFQ-R Cystic Fibrosis Questionnaire-Revised CFTR CF transmembrane conductance regulator protein CFTR CF transmembrane conductance regulator gene CI COFTR CF transmembrane conductance regulator gene CI CRF CSR Clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 CYP cytochrome P450 ECG electroardiogram EDC electroardiogram EDC EENT ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/F heterozygous for the F508del and a minimal function CFTR mutation FFB homozygous for the F508del and a minimal function CFTR mutation FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FDC fixed-dose combination FDC fixed-dose combination FUE 25%-25% Forced expiratory flow, midexpiratory phase FV1 FOC FOC GOA | Abbreviation | Definition |
|---|---|---|
| ALT alanine transaminase AST aspartate transaminase CF cystic fibrosis CFQ-R Cystic Fibrosis Questionnaire-Revised CFTR CF transmembrane conductance regulator protein CFTR CF transmembrane conductance regulator gene CI confidence interval CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 ECG electrocardiogram EDC electronic data capture EENT eyes, cars, nose, and throat ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/MF heterozygous for the F508del and a minimal function CFTR mutation F/S08del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF296-7595 forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Partice Interim analysis ICF informed consent form ICH International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent data monitoring committee IEC independent data monitoring committee IEC independent data monitoring committee IEC independent data monitoring committee IEC independent data monitoring committee | AE | adverse event |
| AST cystic fibrosis CFQ-R cystic Fibrosis Questionnaire-Revised CFTR CF transmembrane conductance regulator protein CFTR CF transmembrane conductance regulator gene CI confidence interval CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 ECG electronic data capture EENT eyes, cars, nose, and throat ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/FF homozygous for the F508del and a minimal function CFTR mutation F/S08del CFTR gene mutation with an in-frame deletion of a phenylalamine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FEF25%-75% forced expiratory flow, midexpiratory phase FEFV <sub>1</sub> forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | ALP | alkaline phosphatase |
| CF cystic fibrosis CFQ-R Cystic Fibrosis Questionnaire-Revised CFTR CF transmembrane conductance regulator protein CFTR CF transmembrane conductance regulator gene CI confidence interval CRF case report form CSR clinical study report CTCAE COmmon Terminology Criteria for Adverse Events CYP cytochrome P450 ECG electrocardiogram EDC electronic data capture EENT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/FF hotomozygous for the F508del and a minimal function CFTR mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FDC fixed-dose combination FE25%,75% FOC and Drug Administration FDC fixed-dose combination FE72-1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMIE International Committee of Medical Journal Editors IDMC independent ethics committee IPD important protocol deviation | ALT | alanine transaminase |
| CFQ-R Cystic Fibrosis Questionnaire-Revised CFTR CF transmembrane conductance regulator protein CFTR CF transmembrane conductance regulator gene CI confidence interval CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 ECG electrocardiogram EDC electronic data capture EENT eyes, cars, nose, and throat ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/MF heterozygous for the F508del and a minimal function CFTR mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FFEF25%-55% forced expiratory flow, midexpiratory phase FEV <sub>1</sub> forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Committee IPD important protocol deviation | AST | aspartate transaminase |
| CFTR CF transmembrane conductance regulator protein CFTR CF transmembrane conductance regulator gene CI confidence interval CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/FF heterozygous for the F508del and a minimal function CFTR mutation CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEV1 forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Committee of Medical Journal Editors IDMC independent ethics committee IEC independent ethics committee IEC independent ethics committee III important protocol deviation | CF | cystic fibrosis |
| CFTR CF transmembrane conductance regulator gene CI confidence interval CRF case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/F heterozygous for the F508del and a minimal function CFTR mutation CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICM International Council for Harmonization ICMJE International Committee of Medical Journal Editors IndMC independent ethics committee IEC independent ethics committee IFD important protocol deviation | CFQ-R | Cystic Fibrosis Questionnaire-Revised |
| CI case report form CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/MF heterozygous for the F508del and a minimal function CFTR mutation F308del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF2394c7594 forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Committee of Medical Journal Editors IDMC independent ethics committee IEC independent ethics committee IPD important protocol deviation | CFTR | CF transmembrane conductance regulator protein |
| CRF clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/MF heterozygous for the F508del and a minimal function CFTR mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF2595-7594 forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | CFTR | CF transmembrane conductance regulator gene |
| CSR clinical study report CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/MF heterozygous for the F508del and a minimal function CFTR mutation CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF2594-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent ethics committee IPD important protocol deviation | CI | confidence interval |
| CTCAE Common Terminology Criteria for Adverse Events CYP cytochrome P450 ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/MF heterozygous for the F508del and a minimal function CFTR mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF25%75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent ethics committee IPD important protocol deviation | CRF | case report form |
| CYP cytochrome P450 ECG electrocardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/MF heterozygous for the F508del and a minimal function CFTR mutation F308del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC fored vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | CSR | clinical study report |
| ECG electroardiogram EDC electronic data capture EENT eyes, ears, nose, and throat ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/MF heterozygous for the F508del and a minimal function CFTR mutation CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF2598-7596 forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent ethics committee IPD important protocol deviation | CTCAE | Common Terminology Criteria for Adverse Events |
| EDC electronic data capture EENT eyes, ears, nose, and throat ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/MF heterozygous for the F508del and a minimal function CFTR mutation CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF125% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent ethics committee IEC indopendent ethics committee IPD important protocol deviation | CYP | cytochrome P450 |
| EENT eyes, ears, nose, and throat ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/MF heterozygous for the F508del and a minimal function CFTR mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent ethics committee IEC independent ethics committee IEC independent ethics committee IPD | ECG | electrocardiogram |
| ETT Early Termination of Treatment EU European Union F/F homozygous for the F508del CFTR mutation F/MF heterozygous for the F508del and a minimal function CFTR mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF2596-7596 forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | EDC | electronic data capture |
| EU European Union F/F homozygous for the F508del CFTR mutation F/MF heterozygous for the F508del and a minimal function CFTR mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IPD important protocol deviation | EENT | eyes, ears, nose, and throat |
| F/F homozygous for the F508del CFTR mutation F/MF heterozygous for the F508del and a minimal function CFTR mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF <sub>25%-75%</sub> forced expiratory flow, midexpiratory phase FEV <sub>1</sub> forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent ethics committee IPD important protocol deviation | ETT | Early Termination of Treatment |
| F/MF heterozygous for the F508del and a minimal function CFTR mutation F508del CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF25%-75% forced expiratory flow, midexpiratory phase FEV1 forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent ethics committee IPD important protocol deviation | EU | European Union |
| CFTR gene mutation with an in-frame deletion of a phenylalanine codon corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF <sub>25%-75%</sub> forced expiratory flow, midexpiratory phase FEV <sub>1</sub> forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent ethics committee IPD important protocol deviation | F/F | homozygous for the F508del CFTR mutation |
| corresponding to position 508 of the wild-type protein FAS Full Analysis Set FDA Food and Drug Administration FDC fixed-dose combination FEF <sub>25%-75%</sub> forced expiratory flow, midexpiratory phase FEV <sub>1</sub> forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | F/MF | heterozygous for the F508del and a minimal function CFTR mutation |
| FDA Food and Drug Administration FDC fixed-dose combination FEF <sub>25%-75%</sub> forced expiratory flow, midexpiratory phase FEV <sub>1</sub> forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IPD important protocol deviation | F508del | |
| FDC fixed-dose combination FEF <sub>25%-75%</sub> forced expiratory flow, midexpiratory phase FEV <sub>1</sub> forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IPD important protocol deviation | FAS | Full Analysis Set |
| FEF <sub>25%-75%</sub> forced expiratory flow, midexpiratory phase FEV <sub>1</sub> forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | FDA | Food and Drug Administration |
| FEV <sub>1</sub> forced expiratory volume in 1 second FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | FDC | fixed-dose combination |
| FSH follicle-stimulating hormone FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | FEF <sub>25%-75%</sub> | forced expiratory flow, midexpiratory phase |
| FVC forced vital capacity GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent ethics committee IEC important protocol deviation | $FEV_1$ | forced expiratory volume in 1 second |
| GCP Good Clinical Practice GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | FSH | follicle-stimulating hormone |
| GGT gamma-glutamyl transferase GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | FVC | forced vital capacity |
| GLI Global Lung Function Initiative GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | GCP | Good Clinical Practice |
| GPS Global Patient Safety HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | GGT | gamma-glutamyl transferase |
| HR heart rate IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | GLI | Global Lung Function Initiative |
| IA interim analysis ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | GPS | Global Patient Safety |
| ICF informed consent form ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | HR | heart rate |
| ICH International Council for Harmonization ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | IA | interim analysis |
| ICMJE International Committee of Medical Journal Editors IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | ICF | informed consent form |
| IDMC independent data monitoring committee IEC independent ethics committee IPD important protocol deviation | ICH | International Council for Harmonization |
| IEC independent ethics committee IPD important protocol deviation | ICMJE | International Committee of Medical Journal Editors |
| IPD important protocol deviation | IDMC | independent data monitoring committee |
| | IEC | independent ethics committee |
| IRB institutional review board | IPD | important protocol deviation |
| | IRB | institutional review board |

IVA ivacaftor

IWRS interactive web response system

LS least squares
LUM lumacaftor
max maximum value

MedDRA Medical Dictionary for Regulatory Activities

min minimum value

MMRM mixed-effects model for repeated measures
OATP1B1/3 organic anion transporting polypeptide 1B1/3

P probability

PD pharmacodynamics
PE physical examination
PEx pulmonary exacerbation

p-gp P-glycoprotein

ppFEV<sub>1</sub> percent predicted forced expiratory volume in 1 second

PR PR interval, segment
PT Preferred Term
q12h every 12 hours
qd once daily

QRS the portion of an ECG comprising the Q, R, and S waves, together representing

ventricular depolarization

QT QT interval

QTcF QT interval corrected by Fridericia's formula

RR interval from the onset of 1 QRS complex to the next; use R-R if using with

"intervals", i.e., "R-R interval"

SAE serious adverse event
SAP statistical analysis plan
SD standard deviation
SOC System Organ Class

SUSAR suspected, unexpected, serious adverse reaction

SwCl sweat chloride
TC triple combination
TE treatment-emergent

TEAE treatment-emergent adverse event

TEZ tezacaftor

ULN upper limit of normal

US United States

#### 5 INTRODUCTION

# 5.1 Background

Cystic fibrosis (CF) is an autosomal recessive chronic disease with serious morbidities and frequent premature mortality. CF affects more than 70,000 individuals worldwide<sup>1</sup> (approximately 30,000 in the US<sup>2</sup> and 45,000 in the EU<sup>3</sup>). Based on its prevalence, CF qualifies as an orphan disease.<sup>4,5</sup>

CF is caused by decreased quantity and/or function of the CFTR protein due to mutations in the *CFTR* gene. CFTR is an ion channel that regulates the flow of chloride and other ions across epithelia in various tissues, including the lungs, pancreas and other gastrointestinal organs, and sweat glands. Decreased CFTR quantity or function results in the failure to regulate chloride transport in these tissues, leading to the multisystem pathology associated with CF. In the lungs, obstruction of airways with thick mucus, establishment of a chronic bacterial infection in the airways, and damaging inflammatory responses are all thought to play a role in causing irreversible structural changes in the lungs, leading to respiratory failure. Progressive loss of lung function is the leading cause of mortality.

The most common disease-causing *CFTR* mutation is F508del, which accounts for approximately 70% of the identified alleles in people with CF. <sup>10</sup> Approximately 40% to 45% of people with CF are homozygous for F508del (F/F), and approximately 85% have at least 1 F508del allele. <sup>2, 3</sup>

Based on the understanding of the molecular defects caused by *CFTR* mutations, 2 complementary approaches have been developed to address the decreased quantity and/or function of CFTR in order to enhance chloride transport in patients with CF. Correctors facilitate the cellular processing and trafficking to increase the quantity of CFTR at the cell surface. Potentiators increase the channel open probability (channel gating activity) of the CFTR protein delivered to the cell surface to enhance ion transport. With differing mechanisms of action, a combination of correctors and potentiators increases F508del CFTR-mediated chloride transport more than either type of modulator alone.

The therapeutic activity of CFTR modulators has been established with products developed by Vertex and approved for the treatment of CF: ivacaftor (IVA) monotherapy (Kalydeco<sup>TM</sup>), lumacaftor (LUM)/IVA (Orkambi<sup>®</sup>), and tezacaftor (TEZ)/IVA (Symdeko<sup>TM</sup>/Symkevi<sup>®</sup>).

VX-445 is a next-generation CFTR corrector. In vitro, the triple combination (TC) of VX-445, TEZ, and IVA (VX-445/TEZ/IVA) increased CFTR chloride transport more than any of the dual combinations (VX-445/TEZ, VX-445/IVA, and TEZ/IVA) or individual components (VX-445, TEZ, and IVA) when added to human bronchial epithelial cells derived from 2 groups of CF patients: those heterozygous for *F508del* with a second *CFTR* allele carrying a minimal function (MF) mutation that is not responsive to TEZ, IVA, and TEZ/IVA (F/MF genotypes); and those homozygous for *F508del* (F/F genotypes).

Additional information about VX-445/TEZ/IVA can be found in the Investigator's Brochure.

## 5.2 Rationale for the Present Study

This study will evaluate the efficacy and safety of VX-445/TEZ/IVA in subjects with CF who have an F/F genotype. The potential for benefit in these patients is supported by in vitro data and

Phase 3 clinical data in subjects with F/F genotypes. In addition, VX-445/TEZ/IVA is generally safe and well tolerated (refer to VX-445 Investigator's Brochure).

The primary endpoint of this study is a widely accepted quality of life measure for subjects with CF; these data are intended to enrich the body of evidence showing that VX-445/TEZ/IVA provides additional benefit to subjects with F/F genotypes over currently available CFTR modulators.

#### 6 STUDY OBJECTIVES

## 6.1 Primary Objective

To evaluate the efficacy of VX-445/TEZ/IVA in CF subjects, homozygous for *F508del* (F/F).

## 6.2 Secondary Objectives

- To evaluate the safety of VX-445/TEZ/IVA
- To evaluate the pharmacodynamics (PD) of VX-445/TEZ/IVA

#### 7 STUDY ENDPOINTS

# 7.1 Primary Endpoint

• Absolute change in CF Questionnaire-Revised (CFQ-R) respiratory domain score from baseline through Week 24

## 7.2 Key Secondary Endpoint

• Absolute change in percent predicted forced expiratory volume in 1 second (ppFEV<sub>1</sub>) from baseline through Week 24

# 7.3 Secondary Endpoints

- Absolute change in sweat chloride (SwCl) from baseline through Week 24
- Safety and tolerability assessments based on adverse events (AEs), clinical laboratory values, ECGs, vital signs, and pulse oximetry

#### 8 STUDY POPULATION

Eligibility will be reviewed and documented by an appropriately qualified member of the investigator's team before subjects receive study drug on Day -28.

Subjects who meet all of the inclusion criteria and none of the exclusion criteria will be eligible.

#### 8.1 Inclusion Criteria

- 1. Subject (or his or her legally appointed and authorized representative) will sign and date an informed consent form (ICF), and, when appropriate, an assent form.
- 2. Willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines, and other study procedures.
- 3. Age 12 years or older, on the date of informed consent.

- 4. Confirmed diagnosis of CF as determined by the investigator.
- 5. Subject has the F/F genotype. Note: If the screening *CFTR* genotype result is not received before Day -28, a previous *CFTR* genotype laboratory report may be used to establish eligibility to enter the Run-in Period. Subjects who have been enrolled and whose screening genotype is not confirmed to be F/F must be discontinued from the study (Section 9.9).
- 6. Forced expiratory volume in 1 second (FEV₁) value ≥40% and ≤90% of predicted mean for age, sex, and height (equations of the Global Lung Function Initiative [GLI])<sup>11</sup> at the Screening Visit. Spirometry measurements must meet American Thoracic Society/European Respiratory Society criteria<sup>12</sup> for acceptability and repeatability.
- 7. Stable CF disease as judged by the investigator.
- 8. Willing to remain on a stable CF treatment regimen (defined in Section 9.5) through completion of study participation.

#### 8.2 Exclusion Criteria

- 1. History of any illness or any clinical condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject. This includes, but is not limited to, the following:
  - Clinically significant cirrhosis with or without portal hypertension.
  - Solid organ or hematological transplantation.
  - Alcohol or drug abuse in the past year, including, but not limited to, cannabis, cocaine, and opiates, as deemed by the investigator.
  - Cancer, except for squamous cell skin cancer, basal cell skin cancer, and Stage 0 cervical carcinoma in situ (all 3 having occurred more than 5 years before screening with no recurrence for the last 5 years).
- 2. Any of the following abnormal laboratory values at screening:
  - Hemoglobin <10 g/dL
  - Total bilirubin  $\ge 2 \times \text{upper limit of normal (ULN)}$
  - Aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT), or alkaline phosphatase (ALP) ≥3 × ULN
  - Abnormal renal function defined as glomerular filtration rate ≤50 mL/min/1.73 m<sup>2</sup> (calculated by the Modification of Diet in Renal Disease Study Equation)<sup>13, 14</sup> for subjects ≥18 years of age and ≤45 mL/min/1.73 m<sup>2</sup> (calculated by the Counahan-Barratt equation)<sup>15</sup> for subjects aged 12 to 17 years (inclusive)
- 3. An acute upper or lower respiratory infection, pulmonary exacerbation(s) (PEx), or changes in therapy (including antibiotics) for sinopulmonary disease within 28 days before the first dose of TEZ/IVA in the Run-in Period (Day -28).
- 4. Lung infection with organisms associated with a more rapid decline in pulmonary status (including, but not limited to, *Burkholderia cenocepacia*, *Burkholderia dolosa*, and *Mycobacterium abscessus*). For subjects who have had a history of a positive culture, the

investigator will apply the following criteria to establish whether the subject is free of infection with such organisms:

- The subject has not had a respiratory tract culture positive for these organisms within the 12 months before the date of informed consent.
- The subject has had at least 2 respiratory tract cultures negative for such organisms within the 12 months before the date of informed consent, with the first and last of these separated by at least 3 months, and the most recent 1 within the 6 months before the date of informed consent.
- 5. An acute illness not related to CF (e.g., gastroenteritis) within 14 days before the first dose of TEZ/IVA in the Run-in Period (Day -28).
- 6. Ongoing or prior participation in a study of an investigational treatment other than a Vertex CFTR modulator within 28 days or 5 terminal half-lives (whichever is longer) before screening. The duration of the elapsed time may be longer if required by local regulations.
- 7. Use of prohibited medications as defined in Table 9-2, within the specified window before the first dose of TEZ/IVA in the Run-in Period (Day -28).
- 8. Pregnant or nursing females. All female subjects must have a negative pregnancy test at Screening/Day -56 (serum test) and TEZ/IVA Run-in Period/Day -28 (urine test).
- 9. The subject or a close relative of the subject is the investigator or a subinvestigator, research assistant, pharmacist, study coordinator, or other staff directly involved with the conduct of the study at that site. However, an adult (aged 18 years or older) who is a relative of a study staff member may be enrolled in the study provided that
  - the adult lives independently of and does not reside with the study staff member, and
  - the adult participates in the study at a site other than the site at which the family member is employed.

#### 9 STUDY IMPLEMENTATION

## 9.1 Study Design

This is a Phase 3, randomized, double-blind, active-controlled, parallel-group, multicenter study (Figure 9-1).



Figure 9-1 Schematic of the Study Design

IVA: ivacaftor; N: number of subjects; TEZ: tezacaftor

Note: The Safety Follow-up Visit is not required for subjects who complete the Week 24 Visit and have enrolled in an open-label study within 28 days after the last dose of study drug.

In the TEZ/IVA Run-in Period, all subjects will receive TEZ 100 mg once daily (qd)/IVA 150 mg every 12 hours (q12h). After completing the TEZ/IVA Run-in Period, subjects will be randomized (1:1) to the TC group or TEZ/IVA group for the Treatment Period. Randomization will be stratified by ppFEV<sub>1</sub> determined during the TEZ/IVA Run-in Period (Day -14 assessment; <70 versus  $\geq$ 70), age at the Screening Visit (<18 versus  $\geq$ 18 years of age), and whether the subject is receiving CFTR modulator treatment at the Screening Visit (yes versus no). If the Day -14 ppFEV<sub>1</sub> value is not valid or not available, the most recent available ppFEV<sub>1</sub> value will be used for stratification.

The dosages for the Treatment Period are shown in Table 9-1.

**Table 9-1** Treatment Period Groups and Dosages

| Treatment Group | VX-445 Dosage | TEZ Dosage | IVA Dosage |
|-----------------|---------------|------------|-------------|
| VX-445/TEZ/IVA | 200 mg qd | 100 mg qd | 150 mg q12h |
| TEZ/IVA | 0 mg qd | 100 mg qd | 150 mg q12h |

IVA: ivacaftor; q12h: every 12 hours; qd: once daily; TEZ: tezacaftor

Note: Study drug administration is described in Section 9.6.

Study visits and assessments to be conducted are shown in Table 3-1 and Table 3-2. All visits will occur within the windows specified.

#### 9.1.1 Screening

The Screening Period will occur within 28 days before the first dose of study drug in the TEZ/IVA Run-in Period.

Screening assessments will be used to confirm that subjects meet the eligibility criteria. The investigator (or an appropriate authorized designee) will obtain informed consent and assent, if applicable, from each subject before any study procedure takes place.

## 9.1.1.1 Repetition of Screening Assessment(s)

Screening assessments may be repeated once to establish study eligibility. If repeat values of the individual assessment(s) are within the eligibility criteria and completed within the screening window, then the subject is eligible for the study.

## 9.1.1.2 Rescreening

Subjects may be rescreened once. If a subject is rescreened, all screening assessments will be repeated, except for:

- *CFTR* genotyping
- Follicle-stimulating hormone (FSH) level (if serum FSH level was in the postmenopausal range as determined by the laboratory performing the test during prior screening)
- Ophthalmologic examination (if performed within 3 months of the date of informed consent, for subjects <18 years of age)

If a subject is rescreened, a new screening window will begin when the first rescreening assessment has been initiated.

## 9.1.1.3 Extension of Screening Period Window

A subject may have the Screening Period window extended by 2 weeks for the following reasons:

- Repetition of the Screening Period assessments (Section 9.1.1.1)
- Unexpected operational or logistic delays, or to meet the eligibility criteria
- Scheduling of ophthalmologic examination (for subjects <18 years of age on the date of informed consent, Section 11.5.6)

## 9.1.2 Tezacaftor/Ivacaftor Run-in Period

The TEZ/IVA Run-in Period has a 4-week duration and is designed to establish a reliable on-treatment (TEZ/IVA) baseline for the Treatment Period. The first dose of open-label TEZ/IVA will be administered at the Day -28 Visit. The last dose of open-label TEZ/IVA will be administered in the evening on Day -1 (1 day before the Day 1 Visit).

The Day -14 spirometry assessment will be used for stratification of randomization to the Treatment Period (Section 9.2).

Subjects who prematurely discontinue study drug treatment during the TEZ/IVA Run-in Period will not be randomized or participate in the Treatment Period (Section 9.1.5.1).

#### 9.1.3 Treatment Period

The Treatment Period will be randomized, double-blind, and active-controlled. It will last approximately 24 weeks (Day 1 to Week 24). Study drug administration details are provided in Section 9.6.

Randomization will occur before the first dose of study drug during the Treatment Period and may occur on either Day -1 or Day 1. Randomization and stratification details are provided in Section 9.2.

To enter the Treatment Period, subjects must have stable CF disease (as judged by the investigator) and have remained on a stable CF treatment regimen during the TEZ/IVA Run-in Period. If these conditions are not met (for example, if the subject has an acute upper or lower respiratory infection, PEx, or changes in therapy [including antibiotics] for sinopulmonary disease within 28 days before the Day 1 Visit [first dose of study drug in the Treatment Period]), subjects may be rescreened once (Section 9.1.1.2) and re-enter the TEZ/IVA Run-in Period on Day -28.

Subjects who prematurely discontinue study drug treatment during the Treatment Period will remain in the study from the time of discontinuation of study drug treatment through the last scheduled study visit and complete the assessments for all study visits, as described in Section 9.1.5.2.

## 9.1.4 Follow-up

The Safety Follow-up Visit will occur approximately  $28 (\pm 7)$  days after the last dose of study drug for subjects who complete study drug dosing and for subjects who prematurely discontinue study drug dosing, as described in Section 9.1.5.

An open-label roll-over study will be available for subjects who complete the Week 24 Visit and are eligible. The Safety Follow-up Visit is not required for subjects who complete the Week 24 Visit and enroll in an open-label roll-over study within 28 days after the last dose of study drug.

## 9.1.5 Early Termination of Treatment

If a subject prematurely discontinues study drug treatment, an Early Termination of Treatment (ETT) Visit should be scheduled as soon as possible after the decision to discontinue treatment. Subjects who prematurely discontinue treatment will also be required to complete the Safety Follow-up Visit, approximately 28 days after their last dose of study drug. The assessments performed at the Safety Follow-up Visit are listed in Table 3-2.

If the ETT Visit occurs 3 weeks or later following the last dose of study drug, then the ETT Visit will replace the Safety Follow-up Visit, and a separate Safety Follow-up Visit will not be required.

If a subject withdraws from the study and also withdraws consent or assent, no further assessments will be performed. Vertex may retain and continue to use any data and samples collected before such withdrawal of consent or assent.

# 9.1.5.1 Discontinuation During the Run-in Period

Subjects who prematurely discontinue study drug treatment during the TEZ/IVA Run-in Period will not be randomized or participate in the Treatment Period. These subjects will complete an ETT Visit and Safety Follow-up Visit (as applicable; see Section 9.1.5). The Safety Follow-up Visit will be their last visit in the study.

## 9.1.5.2 Discontinuation During the Treatment Period

Subjects who prematurely discontinue study drug treatment during the Treatment Period will continue to complete all scheduled study visits following completion of the ETT Visit, as

detailed in Table 3-2. These subjects will complete an ETT Visit and Safety Follow-up Visit (as applicable; see Section 9.1.5).

## 9.1.6 Lost to Follow-up

A subject will be considered lost to follow-up if both of the following occur:

- The subject misses 2 consecutive study visits (telephone contact and/or clinic visit) and is subsequently unable to be contacted by telephone (3 documented attempts by telephone within 2 weeks following the second missed visit).
- The subject does not respond within 2 weeks to a registered letter sent after the 3 attempted telephone contacts.

## 9.1.7 Completion of Study Participation

Completion of study participation for each individual subject is defined as one of the following:

- For subjects who complete the Treatment Period and enter an open-label study within 28 days of the Week 24 Visit: the Week 24 Visit
- For subjects who complete the Treatment Period and do not enter an open-label study within 28 days of the Week 24 Visit: the Safety Follow-up Visit
- For subjects who prematurely discontinue study drug treatment during the Treatment Period but do not withdraw consent (and assent, as applicable): The latest of the Week 24 Visit, ETT Visit, or Safety Follow-up Visit (if required)
- For subjects who prematurely discontinue study drug treatment during the TEZ/IVA Run-in Period but do not withdraw consent (and assent, as applicable): the ETT or Safety Follow-up Visit (if required)
- For subjects who withdraw consent or assent: date of withdrawal of consent or assent, whichever is earlier (Section 9.9)

If subjects are lost to follow-up (Section 9.1.6), the date of completion of study participation will be defined as the date of the last contact.

The end of study is defined in Section 13.2.8.

# 9.2 Method of Assigning Subjects to Treatment Groups

Subjects will be randomized (1:1) to the VX-445/TEZ/IVA or TEZ/IVA group. Randomization will be stratified by ppFEV<sub>1</sub> determined during the TEZ/IVA Run-in Period (Day -14 assessment; <70 versus  $\geq$ 70), age at the Screening Visit (<18 versus  $\geq$ 18 years of age), and whether the subject is receiving CFTR modulator treatment at the Screening Visit (yes versus no). If the Day -14 ppFEV<sub>1</sub> value is not valid or not available, the most recent available ppFEV<sub>1</sub> value will be used for stratification.

An interactive web response system (IWRS) will be used to assign subjects to treatment. The randomization code list will be produced by Vertex Biometrics or a qualified randomization vendor.

## 9.3 Rationale for Study Elements

## 9.3.1 Study Design

A randomized, double-blind, controlled study design was selected to assess the effects of VX-445/TEZ/IVA while avoiding observer bias. TEZ/IVA is considered an appropriate active control since TEZ/IVA (Symdeko/Symkevi) is approved to treat CF in this patient population.

A 4-week TEZ/IVA Run-in Period was incorporated into this study to establish a reliable on-treatment (TEZ/IVA) baseline for comparison during the Treatment Period.

The study will have a 24-week duration to allow for the collection of controlled efficacy and safety data.

The extent of response to CFTR modulator treatment may depend on the subject's ppFEV<sub>1</sub> value (an index of disease severity) before the start of randomized study drug dosing. Some subjects in this study may be receiving treatment with LUM/IVA or TEZ/IVA at screening, while some subjects may not be receiving treatment with CFTR modulators. Therefore, randomization will be stratified by previous CFTR modulator use and ppFEV<sub>1</sub> value determined during the TEZ/IVA Run-in Period after at least 13 days of treatment with TEZ/IVA (Day -14 assessment). Randomization will also be stratified by age at screening. This will ensure a balanced evaluation of adult and adolescent subjects.

## 9.3.2 Study Population

CF patients with the F/F genotype have continuing unmet needs despite the availability of CFTR modulators, and are expected to respond to a TC regimen of VX-445/TEZ/IVA based on results from Phase 2 and Phase 3 studies in this population.

The VX-445 Phases 2 and 3 clinical safety and efficacy data support the enrollment of subjects ≥12 and <18 years of age in this study.

## 9.3.3 Study Drug Dose

#### VX-445 Dosage

A VX-445 dose of 200 mg qd will be administered. This is the dosing regimen that was evaluated in Phase 3 studies of VX-445/TEZ/IVA.

#### **TEZ/IVA Dosage**

TEZ will be administered as 100 mg qd and IVA will be administered as 150 mg q12h. This is the approved dosing regimen for Symdeko/Symkevi.

## 9.3.4 Rationale for Study Assessments

SwCl, spirometry, and CFQ-R endpoints are widely accepted and generally recognized as reliable, accurate, and relevant to the study of individuals with CF and were evaluated in previous registration studies of CFTR modulators.

All safety assessments are standard measurements for clinical studies in drug development.

## 9.4 Study Restrictions

### 9.4.1 Prohibited Medications

Table 9-2 lists prohibited medications. A non-exhaustive list of study prohibitions and cautions for medication will be provided in the Study Reference Manual.

**Table 9-2** Prohibited Medications

| | Timing of Restriction | | |
|---|---|---|---|
| | ~ | End of | - |
| Medication | Start of Restriction | Restriction | Rationale |
| Moderate and strong | None allowed | None allowed | VX-445, TEZ, and IVA are metabolized |
| CYP3A inducers | within 14 days | through | extensively via CYP3A4. Therefore, use of |
| | before the first dose | completion of | moderate and strong inducers of CYP3A and |
| | of the study drug on | study | moderate and strong inhibitors of CYP3A, which |
| | Day -28 | participation | have the potential to alter the exposure of |
| Moderate and strong | None allowed | None allowed | VX-445, TEZ, or IVA, will be prohibited. |
| CYP3A inhibitors | within 14 days | through | |
| (except | before the first dose | completion of | |
| ciprofloxacin)a | of the study drug on | study | |
| | Day -28 | participation | |
| Non-Vertex CFTR | None allowed | None allowed | These agents may confound the results of this |
| modulators | within 28 days or | through | study. |
| (investigational or | 5 terminal half-lives | completion of | |
| approved) | (whichever is | study | |
| | longer) before | participation | |
| | screening | | |
| Vertex CFTR | None allowed from | None allowed | These agents may confound the results of this |
| modulators | the first dose of | until after the last | study. |
| (investigational or | study drug on | dose of study | |
| approved), except | Day -28 | drug | |
| for study drugs | | | |

CYP: cytochrome P450; IVA: ivacaftor; TEZ: tezacaftor

#### 9.5 Prior and Concomitant Medications

Information regarding prior and concomitant medications, including CF medications, other medications, and herbal and naturopathic remedies, will be collected from each subject's source documentation for medications taken within 56 days before the Screening Visit through completion of study participation, as defined in Section 9.1.7.

For subjects who are screened, but are not subsequently randomized into the Treatment Period, details of prior medication will be documented only in the subjects' source documents.

• Subjects should remain on a stable treatment regimen for their CF from 28 days before the TEZ/IVA Run-in Period/Day -28 through completion of study participation. Stable treatment regimen is defined as the current treatment regimen for CF that subjects have been following for at least 28 days before the TEZ/IVA Run-in Period/Day -28. Subjects may remain on Vertex CFTR modulators (investigational or approved) during the Screening Period and may transition directly to the TEZ/IVA Run-in/Day -28 without a washout (Table 9-2). Subjects

<sup>&</sup>lt;sup>a</sup> Ciprofloxacin is not a moderate CYP3A inhibitor on the basis of results of a drug-drug interaction study conducted with IVA, a sensitive CYP3A substrate (Kalydeco [ivacaftor] US Package Insert).

should not initiate long-term treatment with new medication from 28 days before the TEZ/IVA Run-in Period/Day -28 through completion of study participation. Guidelines for stable treatment regimens for CF are as follows:

- o Subjects who are taking inhaled tobramycin or other chronically inhaled antibiotics should remain on that regimen throughout the study.
- o Subjects who cycle onto and off of an inhaled antibiotic should continue on their prior schedule. The timing of the first dose of study drug on the Day 1 Visit should be synchronized as closely as possible (e.g., not more than  $\pm$  3 days) to the first day in the cycle onto the inhaled antibiotic.
- o Subjects who alternate between 2 different inhaled antibiotics should remain on the same cycling schedule during the study. The timing of the first dose of study drug on the Day 1 Visit should be synchronized as closely as possible (e.g., not more than ± 3 days) to the first day in the cycle onto 1 of the inhaled antibiotics.
- Subjects may receive doses of prednisone or prednisolone of up to 10 mg/day chronically, or up to 60 mg daily for up to 5 days.
- VX-445 may inhibit OATP1B1 and OATP1B3, which may increase the exposure of medicinal products that are substrates for these transporters. Substrates such as statins, glyburide, nateglinide, and repaglinide should be used with caution.
- IVA is a weak inhibitor of P-glycoprotein (P-gp). Administration of IVA may increase systemic exposure of medicinal products that are sensitive substrates of P-gp, which may increase or prolong their therapeutic effect and adverse reactions. Digoxin or other substrates of P-gp with a narrow therapeutic index, such as cyclosporine, everolimus, sirolimus, and tacrolimus, should be used with caution and appropriate monitoring.
- IVA may inhibit CYP2C9; therefore during coadministration with warfarin, additional monitoring of the international normalized ratio is recommended. Other medicinal products that are CYP2C9 substrates for which exposure may be increased include glimepiride and glipizide; these should be used with caution.
- Information about bronchodilator use during the study will be collected and documented. Subjects who are using a bronchodilator must have their spirometry assessments performed according to the guidelines provided in Section 11.4.2.

#### 9.6 Administration

### **9.6.1** Dosing

Study drug will be administered orally. All subjects will receive the same number of tablets each day to maintain the blind. Additional information is provided in the Pharmacy Manual.

Study drug should be administered with a fat-containing meal or snack, such as a standard "CF" meal or snack or a standard meal.

- 1. It is recommended that the dose be taken within 30 minutes of the start of the meal or snack.
- 2. Study drug will be administered as fixed-dose combination (FDC) tablet(s) (e.g., 2 VX-445/TEZ/IVA or matching placebo tablets; 1 TEZ/IVA or matching placebo

- tablet) in the morning and as 1 IVA tablet in the evening. For each subject, doses of study drugs should be taken at approximately the same time ( $\pm$  2 hours) each day.
- 3. On days of scheduled visits, the morning dose of study drug will be administered at the site after predose assessments have been completed. A meal or snack will be provided by the site for the morning dose of study drug.
- 4. If a subject's scheduled visit is to occur in the afternoon, the following guidelines must be used:
  - If the dose in the clinic will be within 6 hours of the subject's scheduled morning dose, the subject should withhold their morning dose of study drug and the morning dose will be administered in the clinic.
  - If the dose in the clinic will be more than 6 hours after the subject's scheduled morning dose, the subject should take the morning dose of study drug at home.
- 5. Subjects will be instructed to bring all used and unused materials associated with the study drug to the site; study drug will be dispensed at each visit, as appropriate.

#### 9.6.2 Missed Doses

If 6 hours or less have passed since the missed morning or evening dose, the subject should take the missed dose as soon as possible and continue on the original schedule.

**Morning dose**: If more than 6 hours have passed since the missed morning dose, the subject should take the missed dose as soon as possible and should not take the evening dose.

**Evening dose**: If more than 6 hours have passed since the missed evening dose, the subject should not take the missed dose. The next scheduled morning dose should be taken at the usual time.

Morning and evening doses should not be taken at the same time.

## 9.7 Dose Modification for Toxicity

No dose modifications for toxicity are allowed. Treatment may be interrupted; if any unacceptable toxicity arises, individual subjects will discontinue dosing.

## 9.8 Study Drug Interruption and Stopping Rules

In subjects who have interrupted study drug for >72 hours for any reason, the investigator should resume study drug only after a thorough investigation of the cause for interruption. The investigator should evaluate the subject's clinical stability and only resume drug after the subject is clinically stable and there is no comorbidity or condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.

The medical monitor should be notified of an interruption of study drug that lasts >72 hours for any reason and of the resumption of study drug after such interruption. The medical monitor should be notified of any plan to discontinue study drug.

#### 9.8.1 Liver Function Tests

The central laboratory will notify the medical monitor of instances of ALT or AST  $>3 \times$  ULN in association with total bilirubin  $>2 \times$  ULN that are derived from centrally submitted samples.

Subjects with new treatment-emergent ALT or AST elevations of  $>3 \times ULN$ , with or without total bilirubin  $>2 \times ULN$ , must be followed closely, including confirmatory testing performed by the central laboratory within 48 to 72 hours of the initial finding and subsequent close monitoring of ALT, AST, and bilirubin levels, as clinically indicated.

If a subject cannot return to the site for central laboratory confirmatory testing, a local laboratory may be used. Local laboratory results must be reported immediately to the medical monitor, and the subject must have the tests repeated and sent to the central laboratory as soon as possible (ideally within 48 to 72 hours).

Study drug administration <u>must be interrupted</u> immediately (before confirmatory testing) if any of the following criteria are met:

- ALT or AST  $> 8 \times ULN$
- ALT or AST >5 × ULN for more than 2 weeks
- ALT or AST  $>3 \times$  ULN, in association with total bilirubin  $>2 \times$  ULN and/or clinical jaundice

A thorough investigation of potential causes should be conducted, and the subject should be followed closely for clinical progression.

Study drug administration must be discontinued if the following criterion is met:

• Subsequent ALT or AST values confirm the initial elevation that satisfied the interruption rule (above), and no convincing alternative etiology (e.g., acetaminophen use, viral hepatitis, alcohol ingestion) is identified, regardless of whether transaminase levels have improved

All subjects in whom treatment is discontinued for elevated transaminases (and bilirubin, as applicable) should have these levels monitored closely until levels normalize or return to baseline.

If an alternative, reversible cause of transaminase elevation with or without increased bilirubin or clinical jaundice has been identified, study drug administration may be resumed once transaminases return to baseline or are ≤2 × ULN, whichever is higher. Regardless of the duration of interruption, the medical monitor should be notified before resumption of study drug. Upon resumption of study drug, transaminases and bilirubin should be assessed weekly for 4 weeks. If a protocol-defined transaminase elevation interruption threshold recurs within 4 weeks of rechallenge with the study drug (with confirmation of the initial elevation by repeat testing within 48 to 72 hours), then the study drug must be permanently discontinued, regardless of the presumed etiology.

#### 9.8.2 Rash

Individuals who develop a generalized rash will be monitored closely. Study drug dosing should be interrupted if a subject develops a generalized rash of Grade 3 or higher, or a rash that is considered a serious adverse event (SAE). The investigator will notify the medical monitor of any rash that results in interruption of study drug, is Grade 3 or higher (Section 13.1.1.4), or is an SAE. Investigators should consider additional evaluation including laboratory testing (e.g., complete blood count with differential, liver function tests), photographs of the rash, and dermatology consultation. The investigator may consider resumption of study drug if considered clinically appropriate.

## 9.9 Removal of Subjects

Subjects may withdraw from the study at any time at their own request. Subjects may be withdrawn from study drug treatment at any time at the discretion of the investigator or Vertex for safety, behavior, noncompliance with study procedures, or administrative reasons. If a subject has been withdrawn from study drug treatment, the subject will continue to be followed, provided that the subject has not withdrawn consent (and assent, as applicable).

In addition, a subject must be discontinued from study drug treatment if the subject meets any of the following criteria:

- Has a screening *CFTR* genotype that does not confirm study eligibility if a previous *CFTR* genotype laboratory report was used to establish eligibility. These subjects must be discontinued from the study (Section 8.1)
- Meets any of the stopping (discontinuation) criteria (Section 9.8)
- Becomes pregnant (Section 11.5.7.2)

Subjects who discontinue study drug treatment should return for study assessments, as noted in Section 9.1.5.2.

If a subject does not return for a scheduled visit, reasonable effort will be made to contact the subject. In any circumstance, reasonable effort will be made to document subject outcome. The investigator will inquire about the reason for withdrawal, request that the subject return all unused investigational product(s), request that the subject return for an ETT Visit and Safety Follow-up Visit, if applicable (see Section 9.1.5), and follow up with the subject regarding any unresolved AEs.

If the subject withdraws consent or assent for the study, no further assessments will be performed. Vertex may retain and continue using the study data and samples after the study is over, and may use the samples and information in the development of the study compound, and for other drugs and diagnostics, in publications and presentations, and for education purposes. If the subject withdraws from the study, the study data and samples collected will remain part of the study. A subject will not be able to request the withdrawal of his/her information from the study data. A subject may request destruction of the samples collected from him/her during the study as long as those samples can be identified as his/her samples.

## 9.10 Replacement of Subjects

Subjects who withdraw or are withdrawn before the first dose of randomized study drug on Day 1 of the Treatment Period may be replaced.

Subjects who withdraw or are withdrawn for nonsafety reasons during the study drug treatment periods may be replaced at Vertex's discretion.

#### 10 STUDY DRUG INFORMATION AND MANAGEMENT

During the TEZ/IVA Run-in Period, study drug refers to TEZ/IVA and IVA.

During the Treatment Period, study drug refers to VX-445/TEZ/IVA and matching placebo, TEZ/IVA and matching placebo, and IVA.

## 10.1 Preparation and Dispensing

Study drug may be dispensed only under the supervision of the investigator or an authorized designee and only for administration to the study subjects.

## 10.2 Packaging and Labeling

Study drug tablets will be supplied in blister cards by Vertex. Study drug labeling will be in compliance with applicable local and national regulations. Additional details regarding packaging, labeling, and dispensing for study drug will be in the Pharmacy Manual.

## 10.3 Study Drug Supply, Storage, and Handling

VX-445/TEZ/IVA will be supplied as FDC film-coated tablets containing 100 mg VX-445, 50 mg TEZ, and 75 mg IVA. Matching VX-445/TEZ/IVA placebo tablets will be of similar size and appearance and contain 0 mg VX-445, 0 mg TEZ, and 0 mg IVA (Table 10-1).

TEZ/IVA will be supplied as FDC film-coated tablets containing 100 mg TEZ and 150 mg IVA. A matching TEZ/IVA placebo tablet will be of similar size and appearance and contain 0 mg TEZ and 0 mg IVA (Table 10-1).

IVA will be supplied as a film-coated tablet containing 150 mg IVA (Table 10-1).

Blister cards must be stored under conditions noted in the Pharmacy Manual. The investigator, or an authorized designee (e.g., a licensed pharmacist), will ensure that all investigational product is stored in a secured area, under recommended storage conditions, and in accordance with applicable regulatory requirements. To ensure adequate records, all study drugs will be accounted for via the drug accountability forms as instructed by Vertex.

Table 10-1 Study Drug: Strength/Dosing Form/Route

| Drug Name, Dosing Form, Route | Strength |
|-----------------------------------------------|----------|
| VX-445/TEZ/IVA, FDC tablet, oral | |
| VX-445 | 100 mg |
| TEZ | 50 mg |
| IVA | 75 mg |
| VX-445/TEZ/IVA-matching placebo, tablet, oral | 0 mg |
| TEZ/IVA, FDC tablet, oral | |
| TEZ | 100 mg |
| IVA | 150 mg |
| TEZ/IVA-matching placebo, tablet, oral | 0 mg |
| IVA, tablet, oral | 150 mg |

FDC: fixed-dose combination; IVA: ivacaftor; TEZ: tezacaftor

## 10.4 Drug Accountability

The pharmacist or designated study site staff will maintain information regarding the dates and amounts of (1) study drug received; (2) study drug dispensed to the subjects; and (3) study drug returned by the subjects. Subjects will be instructed to return all used and unused materials associated with the study drug to the site. These materials will be retained at the site according to instructions provided by Vertex or its designee. The study monitor will review study drug records and inventory throughout the study.

If a site uses a site-specific drug accountability system and/or process, including processes associated with the destruction of returned materials, the process must be documented and approved by Vertex. The study monitor must review the drug accountability documentation on a regular basis. The study monitor will promptly communicate to Vertex any discrepancies he/she is unable to resolve with the site.

## 10.5 Disposal, Return, or Retention of Unused Drug

The study site staff or pharmacy personnel will retain all materials returned by the subjects until the study monitor has performed drug accountability. The investigator will ensure that the materials are destroyed in compliance with applicable environmental regulations, institutional policy, and any special instructions provided by Vertex. Destruction will be adequately documented.

## 10.6 Compliance

To ensure treatment compliance, the investigator or designee will supervise all study drug dosing that occurs at the site. At each visit, site personnel will review that the subject is compliant with study drug dosing and remind the subject of study drug dosing requirements. Compliance will also be assessed by ongoing study drug count.

If a subject demonstrates continued noncompliance of study drug dosing despite educational efforts, the investigator should consider discontinuing the subject from the study.

## 10.7 Blinding and Unblinding

This will be a double-blind study.

## 10.7.1 Blinding

All subjects (and their parents/caregivers/companions), site personnel (including the investigator, the site monitor, and the study team), and members of the Vertex study team will be blinded to the treatment codes.

Individuals who may be unblinded include only the following:

- Any site personnel for whom this information is important to ensure the safety of the subject in the event of a life-threatening medical emergency
- Any site personnel for whom this information is important to ensure the safety of the subject and her fetus in the event of a pregnancy
- Vertex Global Patient Safety (GPS) and Regulatory Affairs personnel to satisfy SAE processing and reporting regulations
- Vendor preparing the final (production) randomization list
- Vertex IWRS Manager
- Vertex Clinical Supply Chain

A limited Vertex team may be unblinded if an interim analysis (IA) is performed. Members of the limited Vertex unblinded team will not be involved in or influence the conduct of the remaining part of the study to protect the integrity of the study (Section 12.3.5.1).

## Access to Spirometry and SwCl Results:

During the conduct of the study, the Vertex study team will not have access to the spirometry or SwCl results after the first dose of study drug in the Treatment Period.

Shortly before any planned efficacy analysis is conducted, the spirometry and SwCl data will be reviewed for data cleaning purposes by a biostatistician who does not have access to the treatment codes.

Individual SwCl test results will not be disclosed to the study sites with the exception of the screening values. Subjects and their parents/caregivers/companions should not be informed of study-related spirometry results until Vertex has determined that the study has completed (i.e., clinical study report [CSR] finalization), regardless of whether the subject has prematurely discontinued treatment.

## 10.7.2 Unblinding

At the initiation of the study, study site personnel will be instructed on the method for breaking the blind. The unblinding method will be either manual or electronic.

# **Unblinding of Individual Subject Treatment Assignments by Investigator for Medical Emergencies or Urgent Clinical Situations**

Unblinding of the individual subject's treatment by the investigator will be limited to medical emergencies or urgent clinical situations in which knowledge of the subject's study treatment is necessary for clinical management. In such cases, investigators will use their best judgment as to whether to unblind without first attempting to contact the medical monitor to discuss unblinding. If investigators deem it unnecessary to unblind immediately, they will first attempt to contact the medical monitor to discuss unblinding. If investigators have tried but are unable to reach the medical monitor, they will use their best judgment, based on the nature and urgency of the clinical situation, and may proceed with unblinding.

Contact information for the medical monitor (or appropriate backup) will be in a separate document.

If a subject's treatment assignment has been unblinded for a medical emergency or urgent clinical situation, the medical monitor will be notified within 24 hours of the unblinding event. The reason and the date of the unblinding will be documented clearly in the subject's study file. Information about the treatment assignment obtained from the unblinding will be maintained in a secure location with controlled access and will not be shared with Vertex, the contract research organization, or any site personnel (other than the physician treating the subject). In addition, the investigator will consider whether the clinical event that prompted unblinding will be considered an SAE, according to the regulatory definitions or criteria for SAEs, and if so, submit an SAE report to Vertex GPS or designee, per Section 13.1.2.

# **Unblinding of Individual Subject Treatment Assignments by Vertex GPS or Designee for SAEs or Safety Concerns**

Vertex GPS or designee will also unblind any SAE reports in compliance with regulatory reporting requirements. In addition, Vertex may, for matters relating to safety, unblind individual subjects at any time.

## **Unblinding: Interim Analysis**

A limited Vertex team may be unblinded if an IA is performed. Members of the limited Vertex unblinded team will not be involved in or influence the conduct of the remaining part of the study to protect the integrity of the study (Section 12.3.5.1). Regardless of the outcome of the IA, subjects (and their parents/caregivers/companions), site personnel (including the investigator, the site monitor, and the study team), and members of the Vertex study team will remain blinded until the final database lock.

#### 11 ASSESSMENTS

## 11.1 Timing of Assessments

The timing of assessments is shown in Table 3-1 and Table 3-2.

## 11.2 Subject and Disease Characteristics

Subject and disease characteristics include the following: demographics, medical history, height, and weight.

Medical history will be elicited from each subject and extracted from medical records during screening. Based on the medical history, the subject will be assessed for any disqualifying medical conditions as specified in the inclusion and exclusion criteria. The medical history will include a complete review of systems, medical and surgical histories, and any allergies.

## 11.3 Pharmacodynamics: Sweat Chloride

SwCl samples will be collected with an approved collection device. Each collection will occur before study drug dosing (Section 9.6.1). At each time point, 2 samples will be collected, 1 from each arm (left and right). Sweat samples will be sent to a central laboratory for testing and interpretation of results. Specific instructions for the collection, handling, processing, and shipping of SwCl samples to the central laboratory will be provided separately.

See Section 10.7.1 for information about access to SwCl results.

## 11.4 Efficacy

# 11.4.1 Cystic Fibrosis Questionnaire-Revised

The questionnaires provide information about demographics; general quality of life, school, work, or daily activities; and symptom difficulties (pertaining to CF).

Subjects will be asked to complete the CFQ-R in their native language, if validated translations are available. <sup>16, 17</sup> If there is no validated translation available in the subject's native language, the subject will not complete the questionnaire. Copies of the CFQ-R used will be provided in the Study Reference Manual. Validated translations of the CFQ-R, if available, will be provided for participating centers in non-English-speaking countries. <sup>18, 19</sup>

The CFQ-R will be completed before any other assessments (except signing of ICF) are performed at that visit.

Subjects who are 12 and 13 years of age at the date of informed consent will complete the CFQ-R Child version themselves, and their parents/caregivers will complete the CFQ-R Parent version, at all visits, regardless of whether the subject subsequently turns 14 years of age during the study. Subjects 14 years of age and older at the date of informed consent will complete the Adolescent/Adult version of the questionnaire themselves at all visits.

## 11.4.2 Spirometry

Spirometry will be performed according to the American Thoracic Society Guidelines/European Respiratory Society Guidelines<sup>12</sup> and according to the additional guidelines that follow.

Pre-bronchodilator spirometry is defined as spirometry testing performed for subjects who have

- withheld their short-acting bronchodilators (e.g., albuterol) or anticholinergic (e.g., ipratropium bromide [Atrovent<sup>®</sup>]) for more than 4 hours before the spirometry assessment;
- withheld their long-acting bronchodilator (e.g., salmeterol) for more than 12 hours before the spirometry assessment; and
- withheld their once-daily, long-acting bronchodilator (e.g., tiotropium bromide [Spiriva®]) for more than 24 hours before the spirometry assessment.

During the Screening Period, spirometry assessments may be performed pre- or post-bronchodilator. At all other visits, all spirometry assessments should be performed pre-bronchodilator. During the Treatment Period, spirometry assessments must be performed before study drug dosing (Section 9.6.1) at approximately the same time at each visit. In the event that a subject forgets to withhold bronchodilator(s), spirometry should be performed according to the following:

- If a subject's Day 1 spirometry assessment is pre-bronchodilator but, on a subsequent visit, the subject forgets to withhold bronchodilator use, a post-bronchodilator spirometry assessment will be obtained for that visit only, and the visit will not be rescheduled.
- If, on Day 1, the subject forgets to withhold his/her dose of bronchodilator, spirometry should be performed post-bronchodilator, and all subsequent spirometric measurements (according to the schedule of assessments in Table 3-2) should be performed post-bronchodilator.
- Each spirometry assessment will be recorded in the source documents as pre- or post-bronchodilator.

All sites will be provided with spirometers to be used for all study assessments. Spirometry data will be transmitted to a centralized spirometry service for quality review. The investigator's assessment of the spirometry results will be used for the screening assessment and determination of eligibility.

See Section 10.7.1 for information about access to spirometry results.

The measured spirometric values listed below will be converted to percent predicted values using the standard equations of GLI.<sup>11</sup>

- FEV<sub>1</sub> (L)
- Forced vital capacity (FVC) (L)
- FEV<sub>1</sub>/FVC (ratio)
- Forced expiratory flow, midexpiratory phase (FEF<sub>25%-75%</sub>) (L/s)

## 11.4.3 Height and Weight

Height and weight will be measured with shoes off. Following screening, height will be collected only for subjects  $\leq$ 21 years of age on the date of informed consent.

#### 11.5 Safety

Safety evaluations will include AEs, clinical laboratory assessments, and clinical evaluation of vital signs, ECGs, physical examinations (PEs), and pulse oximetry.

For subjects <18 years of age on the date of informed consent, ophthalmological examinations will also be performed at screening (if not done within preceding 3 months) and at Week 24 (or ETT Visit or Safety Follow-up Visit).

#### 11.5.1 Adverse Events

All AEs will be assessed, documented, and reported in accordance with ICH GCP guidelines. Section 13.1 outlines the definitions, collection periods, criteria, and procedures for documenting, grading, and reporting AEs. A separate document that details AE case report form (CRF) completion guidelines for investigators as well as training will be provided.

## 11.5.2 Clinical Laboratory Assessments

Blood and urine samples will be analyzed at a central laboratory, with the exception of the urine pregnancy tests. As described below, urine pregnancy tests will either be analyzed by the site or at home using a home kit. On Day 1, blood samples will be collected before the first dose of the study drug.

Laboratory test results that are abnormal and considered clinically significant will be reported as AEs.

The safety laboratory test panels are shown in Table 11-1.

**Table 11-1** Safety Laboratory Test Panels

| Serum Chemistry | Hematology | Urinalysis <sup>a</sup> |
|---|---|---|
| Glucose | Hemoglobin | Leukocyte esterase |
| Blood urea nitrogen <sup>b</sup> | Erythrocytes | Nitrite |
| Creatinine | Mean corpuscular volume | Urobilinogen |
| Sodium | Platelets | Urine protein |
| Potassium | Reticulocytes | pН |
| Calcium | Leukocytes | Urine blood |
| Chloride | Differential (absolute and percent): | Specific gravity |
| Magnesium | Eosinophils | Urine ketones |
| Bicarbonate | Basophils | Urine bilirubin |
| Inorganic phosphate | Neutrophils | Urine glucose |
| Total and direct bilirubin | Lymphocytes | |
| Alkaline phosphatase | Monocytes | |
| Aspartate transaminase | Coagulation Studies | |
| Alanine transaminase | Activated partial thromboplastin time | |
| Amylase | Prothrombin time | |
| Lipase | Prothrombin time International | |
| Gamma-glutamyl transferase | Normalized Ratio | |
| Protein | | |
| Albumin | | |
| Creatine kinase | | |
| Total cholesterol | | |
| Lactate dehydrogenase | | |

Note: Haptoglobin may be analyzed if judged to be clinically appropriate by the investigator.

Pregnancy (β-human chorionic gonadotropin) Tests for female subjects: All female subjects must have a serum pregnancy test at screening. Serum pregnancy tests will be performed at the study site and analyzed at the central laboratory. Urine pregnancy tests will either be performed and analyzed at the site or, when there is no clinic visit scheduled, at home by using a home kit provided by the site. Results will be reported to the site by telephone. The urine pregnancy test on Day 1 must be negative before the first dose of study drug. Additional pregnancy tests may be required according to local regulations and/or requirements.

<u>FSH</u>: Blood samples for FSH will be measured as needed for any suspected postmenopausal female with at least 12 months of continuous spontaneous amenorrhea. Serum FSH levels must be in the postmenopausal range as determined by the laboratory performing the test.

<u>CFTR</u> Genotype (Screening Period Only): CFTR genotyping will be performed for all subjects. If the screening CFTR genotype result is not received before randomization, a previous CFTR genotype laboratory report may be used to establish eligibility. Subjects who have been randomized and whose screening genotype does not confirm study eligibility must be discontinued from the study (Section 9.9).

<u>Additional Evaluations</u>: Additional clinical laboratory evaluations will be performed at other times if judged to be clinically appropriate.

If urinalysis results are positive for leukocyte esterase, nitrite, protein, or blood, microscopic examination of urine will be performed, and results will be provided for leukocytes, erythrocytes, crystals, bacteria, and casts.

If blood urea nitrogen cannot be collected, urea may be substituted.
For the purposes of study conduct and unless noted otherwise, only laboratory tests done in the central laboratory may be used. Local laboratories may be used at the discretion of the local investigator for management of urgent medical issues. If a local laboratory test value is found to be abnormal and clinically significant, it will be verified by the central laboratory as soon as possible after the investigator becomes aware of the abnormal result. If it is not possible to send a timely specimen to the central laboratory (e.g., the subject was hospitalized elsewhere), the investigator may base the assessment of an AE on the local laboratory value.

## 11.5.3 Physical Examinations and Vital Signs

A PE of all body systems and vital signs assessments will be performed at screening and select study visits (see Table 3-1 and Table 3-2). At other visits, symptom-directed PEs and symptom-directed vital sign assessments will occur at any time if deemed necessary by the investigator or healthcare provider.

A complete PE includes a review of the following systems: head, neck, and thyroid; eyes, ears, nose, and throat (EENT); respiratory; cardiovascular; lymph nodes; abdomen; skin; musculoskeletal; and neurological. Breast, anorectal, and genital examinations will be performed when medically indicated. After screening, any clinically significant abnormal findings in PEs will be reported as AEs.

Vital signs include blood pressure (systolic and diastolic), temperature, pulse rate, and respiration rate. These will be assessed before dosing and following at least a 5-minute rest. A consistent methodology should be used for repeat measurements of these parameters at a clinical site.

## 11.5.4 Pulse Oximetry

Pulse oximetry is a noninvasive measure of oxygen delivery to the tissues and has been correlated with clinical status and lung function. Arterial oxygen saturation by pulse oximetry will be assessed following at least a 5-minute rest and before study drug dosing. At visits when study drug is taken at the site, pulse oximetry will be collected before study drug dosing (Section 9.6.1).

## 11.5.5 Electrocardiograms

Standard 12-lead ECGs will be performed using a machine with printout according to the schedule of assessments (Table 3-1 and Table 3-2). Additional standard 12-lead ECGs will be performed at any other time if clinically indicated. Subjects will be instructed to rest for at least 5 minutes before having an ECG performed.

The ECG traces will be manually read at the study site. A printout of the ECG traces will be made for safety review by the investigator and maintained with source documentation. Clinically significant ECG abnormalities occurring during the study through completion of study participation will be recorded as AEs.

To ensure the safety of the subjects, a qualified individual at the study site will make comparisons to baseline measurements. If the QTcF is increased by >60 msec from the baseline or an absolute QTcF value is ≥500 msec for any scheduled ECG, 2 additional ECGs will be performed approximately 2 to 4 minutes apart to confirm the original measurement. If either of the QTcF values from these repeated ECGs remains above the threshold value (>60 msec from baseline or ≥500 msec), a single ECG will be repeated at least hourly until QTcF values from

2 successive ECGs fall below the threshold value that triggered the repeat measurement. Further details pertaining to ECGs will be provided to sites in the ECG Manual.

## 11.5.6 Ophthalmologic Examination

Ophthalmologic examinations will be conducted only for subjects who are <18 years of age on the date of informed consent. The examination does not need to be completed if there is documentation of bilateral lens removal for the subject.

All examinations will be conducted by a licensed ophthalmologist or optometrist and will include:

- measurement of best-corrected distance visual acuity of each eye; and
- pharmacologically-dilated examination of the lens with a slit lamp

The screening examination does not need to be conducted if there is documentation of an examination meeting the protocol requirements that was conducted within 3 months before the date of informed consent.

In addition to the screening ophthalmologic examination, subjects who are <18 years of age on the date of informed consent and who have completed at least 12 weeks of study drug treatment will have a single ophthalmologic examination at either the ETT or Week 24 Visit (whichever comes first), except for those subjects who have withdrawn consent or assent. This examination should be completed within 4 weeks before the Week 24 Visit, unless the subject prematurely discontinues study drug, in which case this examination should occur by the Safety Follow-up Visit (or ETT Visit for subjects who do not complete a Safety Follow-up Visit), as described in Table 3-2.

Any clinically significant abnormal findings will be reported as AEs.

### 11.5.7 Contraception and Pregnancy

The effects of VX-445 monotherapy or in combination with TEZ/IVA on conception, pregnancy, and lactation in humans are not known. VX-445, TEZ, and IVA did not show genotoxic potential in a standard battery of in vitro (Ames test, chromosomal aberration, or micronucleus in cultured mammalian cells) and in vivo (rodent micronucleus) studies. Reproductive toxicology studies of VX-445, TEZ, and IVA have not shown teratogenicity in rats and rabbits.

## 11.5.7.1 Contraception

### Contraception requirement for a couple is waived for the following:

- True abstinence for the subject, when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception. True abstinence must be practiced from the Screening Visit through 90 days after the last dose of study drug.
- If the male is infertile (e.g., bilateral orchiectomy). If a male subject is assumed to have complete bilateral absence of the vas deferens, infertility must be documented before the first dose of study drug (e.g., examination of a semen specimen or by demonstration of the absence of the vas deferens by ultrasound).
- If the female is of non-childbearing potential. To be considered of non-childbearing potential, the female must meet at least 1 of the following criteria:

- o Postmenopausal: Amenorrheic for at least 12 consecutive months and a serum FSH level within the laboratory's reference range for postmenopausal females
- o Documented hysterectomy or bilateral oophorectomy/salpingo-oophorectomy

Note: All other females (including females with tubal ligations and pre-menarchal females) will be considered to be of childbearing potential.

• Same-sex relationships

For subjects for whom the contraception requirement is not waived, study participation requires a commitment from the subject that at least 1 acceptable method of contraception is used as a couple. Methods of contraception must be in successful use from signing of consent, approximately 28 days before the first dose of study drug (unless otherwise noted), and until 90 days following the last dose of study drug. Additional contraception requirements may need to be followed according to local regulations and/or requirements. Acceptable methods of contraception are listed in Table 11-2.

**Table 11-2** Acceptable Methods of Contraception

| | Male Subjects and Their<br>Female (Non-study)<br>Partners | Female Subjects and<br>Their Male (Non-study)<br>Partners |
|---|---|---|
| Vasectomy performed at least 6 months previously, with a documented negative postvasectomy semen analysis for sperm | Yes | Yes |
| Bilateral tubal occlusion (e.g., ligation) performed at least 6 months previously | Yes | Yes |
| Male or female condom with or without spermicide <sup>a</sup> | Yes | Yes |
| Female barrier contraception (such as diaphragm, cervical cap, or sponge) with spermicide | Yes | Yes |
| Continuous use of an intrauterine device for at least 90 days before the first dose of study drug | | |
| Hormone-releasing | Yes | Yes |
| Non-hormone releasing | Yes | Yes |
| Oral, implanted, injected, or vaginal hormonal contraceptives, if successfully used for at least 60 days before the first dose of study drug | Yes | Yes |

<sup>&</sup>lt;sup>a</sup> A female condom cannot be used with a male condom due to risk of tearing.

### **Additional notes:**

- If over the course of the study, the subject meets the criteria for waiving the contraception requirements, the subject does not need to follow the contraceptive methods listed in Table 11-2.
- If, over the course of the study, the subject's status changes and the subject does not meet the criteria for waiving the contraception requirements, the subject must begin following the contraceptive methods listed in Table 11-2.
- Male subjects must not donate sperm during the period starting from the first dose of study drug until 90 days after the last dose of study drug.

- Female subjects should not nurse a child during the period starting from the first dose of study drug until 90 days after the last dose of study drug.
- For male subjects with a female partner of childbearing potential, the couple should not plan to become pregnant during the study or within 90 days after the last dose of study drug, with the exception of couples who plan to become pregnant by artificial insemination using sperm banked by the male subject before the first dose of study drug or sperm from another source.

## 11.5.7.2 **Pregnancy**

Subjects will be counseled to inform the investigator of any pregnancy that occurs during study treatment and for 90 days after the last dose of study drug.

If a female subject becomes pregnant during study participation, study drug will be permanently discontinued immediately. The investigator will notify the medical monitor and Vertex GPS within 24 hours of the site's knowledge of the subject's (or partner's) pregnancy using the Pregnancy Information Collection Form. Male subjects with female partners who become pregnant during the study must use a male condom to avoid exposure of a potential embryo or fetus to study drug via the seminal fluid.

If confirmed to be on active drug, the subject or partner will be followed until the end of the pregnancy and the infant will be followed for 1 year after the birth, provided informed consent (and assent, as applicable) is obtained. A separate ICF will be provided to explain these follow-up activities. Pregnancy itself does not constitute an AE.

### 12 STATISTICAL AND ANALYTICAL PLANS

This section presents a summary of the planned analyses for this protocol. Statistical analysis details will be provided in the statistical analysis plan (SAP), which will be finalized before the clinical data lock for the study and treatment unblinding.

## 12.1 Sample Size and Power

Up to approximately 158 subjects will be enrolled and randomized (1:1) to the VX-445/TEZ/IVA group or the TEZ/IVA group. Information regarding the powering of primary and key secondary endpoints is provided below.

### **Power for Primary Efficacy Endpoint**

The primary efficacy endpoint is the absolute change in CFQ-R respiratory domain score from baseline through Week 24. The primary null hypothesis to be tested is that the mean absolute change in CFQ-R respiratory domain score from baseline is the same for the 2 treatment groups, VX-445/TEZ/IVA and TEZ/IVA. The null hypothesis will be tested at a 2-sided significance level of 0.05.

Assuming a within-group SD of 18 and a treatment difference of 10 between VX-445/TEZ/IVA and TEZ/IVA, a sample size of 71 subjects completing the Treatment Period in each group for a total of 142 subjects will have approximately 90% power for the CFQ-R respiratory domain score hypothesis testing, based on a 2-sample t-test at a significance level of 0.05 (2-sided). Assuming a 10% dropout rate, up to approximately 158 subjects will be enrolled.

## **Power for Key Secondary Endpoint**

The key secondary endpoint is the absolute change in ppFEV<sub>1</sub> from baseline through Week 24. Assuming a within-group SD of 7 percentage points and a treatment difference of 5 between VX-445/TEZ/IVA and TEZ/IVA, a sample size of 71 subjects completing the Treatment Period in each group for a total of 142 subjects will have approximately 98% power for the ppFEV1 hypothesis testing, based on a 2-sample t-test at a significant level of 0.05 (2-sided). Assuming a 10% dropout rate, approximately 158 subjects will be enrolled.

All power calculations were based on EAST software Version 6.4.

## 12.2 Analysis Sets

The following analysis sets are defined: All Subjects Set, Full Analysis Set (FAS), and Safety Set. Additional analysis sets related to the Run-in Period will be defined in the SAP, as appropriate.

The **All Subjects Set** will include all subjects who were randomized or received at least 1 dose of study drug. This analysis set will be used for all individual subject data listings and disposition summary tables, unless otherwise specified.

The **FAS** will include all randomized subjects who carry the intended *CFTR* allele mutation and receive at least 1 dose of study drug in the Treatment Period. The FAS will be used to summarize subject demographics and baseline characteristics, and for all efficacy analyses in which subjects will be analyzed according to their randomized treatment group, unless otherwise specified.

The **Safety Set for the Treatment Period** will include all subjects who receive at least 1 dose of study drug in the Treatment Period. This safety set will be used for all safety analyses in which subjects will be analyzed according to the treatment they receive, unless otherwise specified.

The **Safety Set for the Run-in Period** will include all subjects who received at least 1 dose of study drug in the Run-in Period.

## 12.3 Statistical Analysis

### 12.3.1 General Considerations

Continuous variables will be summarized using the following descriptive summary statistics: the number of subjects (n), mean, SD, median, minimum value (min), and maximum value (max).

Categorical variables will be summarized using counts and percentages.

The **baseline value**, unless otherwise specified, will be defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of study drug in the Treatment Period (i.e., the Day 1 Visit). For ECG, baseline will be defined as the most recent pretreatment measurement (or the average of triplicate measurements, if the most recent pretreatment measurement is obtained in triplicate) before the first dose of study drug in the Treatment Period (i.e., the Day 1 Visit).

**Absolute change** from baseline will be calculated as post-baseline value – baseline value.

The Treatment-emergent (TE) Period for the Run-in Period will be from the first dose of study drug in the Run-in Period to (1) the first dose of study drug in the Treatment Period for subjects who complete the Run-in Period and continue to the Treatment Period, or (2) 28 days

after the last dose date of study drug in the Run-in Period for subjects who do not continue to the Treatment Period (e.g., subjects who do not meet the conditions to enter the Treatment Period).

The **TE Period for the Treatment Period** will include the time from the first dose date of study drug in the Treatment Period (VX-445/TEZ/IVA or placebo + TEZ/IVA) to 28 days after the last dose of the study drug or to the completion of study participation date (as defined in Section 9.1.7), whichever occurs first.

## 12.3.2 Background Characteristics

## 12.3.2.1 Subject Disposition

The number and percentage of subjects in each disposition category (e.g., randomized, included in the FAS, included in the Safety Set, completed Treatment Period, completed study, prematurely discontinued treatment or study with a breakdown of the reasons for discontinuation, and entered an open-label study) will be summarized overall and by treatment group.

An additional subject disposition summary related to the TEZ/IVA Run-in Period will be defined in the SAP, as appropriate.

### 12.3.2.2 Demographics and Baseline Characteristics

Demographic, medical history, and baseline characteristics will be summarized using descriptive summary statistics.

The following demographics and baseline characteristics will be summarized overall and by treatment group for the FAS, and will include (but are not limited to): sex, race, age, baseline weight, baseline height, baseline body mass index, baseline CFQ-R, baseline ppFEV<sub>1</sub>, and baseline SwCl.

Medical history will be summarized by MedDRA System Organ Class (SOC) and Preferred Term (PT) for the FAS.

### 12.3.2.3 Prior and Concomitant Medications

Medications will be coded using the World Health Organization Drug-Dictionary and categorized as follows:

- **Prior medication**: any medication that was administered during the 56 days before the first dose of study drug in the Treatment Period but not in the Run-in Period. For subjects who discontinue during the Run-in Period and whose first dose of study drug in the Treatment Period is not available, prior medication will be any medication that was administered during the 56 days before the last dose of study drug in the Run-in Period but before the first dose in the Run-in Period
- Concomitant medication during the Run-in Period: medication continued or newly received during the TE Period for the Run-in Period
- Concomitant medication during the Treatment Period: medication continued or newly received during the TE Period for the Treatment Period
- Post-treatment medication: medication continued or newly received after:

- o the TE Period for the Run-in Period if the subject did not receive study drug in the Treatment Period
- o the TE Period for the Treatment Period for subjects who received study drug in the Treatment Period

A given medication may be classified as a prior medication, a concomitant medication, or a post-treatment medication; both prior and concomitant; both concomitant and post-treatment; or prior, concomitant, and post-treatment. If a medication has a missing or partially missing start/end date or time and if it cannot be determined whether it was taken before the first dose of study drug, concomitantly during the TE Period, or after the TE Period, it will be considered in all 3 categories of prior, concomitant, and post-treatment medication.

Prior medications and concomitant medications will be summarized descriptively by Preferred Name based on the FAS. Post-treatment medications will be provided separately in an individual subject data listing.

## 12.3.2.4 Study Drug Exposure and Compliance

Study drug exposure and compliance will be summarized for the Treatment Period only.

Study drug exposure will be summarized overall and by treatment group, based on the Safety Set in terms of the duration of treatment a subject received (in days), defined as the last day – the first day of study drug plus 1, regardless of study drug interruption.

Study drug compliance will be summarized overall and by treatment group based on the FAS, and will be calculated as:  $100 \times [1$ - (total number of days of study drug interruption) / (duration of study drug exposure in days)]. A study drug interruption on a given day is defined as an interruption of any study drug on that day.

### 12.3.2.5 Important Protocol Deviations

An important protocol deviation (IPD) is a deviation that may significantly affect the completeness, accuracy, or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being. The rules for identifying an IPD will be described in the SAP.

All IPDs will be provided in an individual subject data listing and summarized, as appropriate.

### 12.3.3 Efficacy and Pharmacodynamic Analyses

The primary objective of the study is the evaluation of the efficacy of VX-445/TEZ/IVA. The analysis in this section will be based on the FAS, unless otherwise specified.

## 12.3.3.1 Analysis of Primary Endpoint

The primary efficacy endpoint is the **absolute change in CFQ-R respiratory domain score from baseline through Week 24**. The analysis of this endpoint will be performed using a mixed-effects model for repeated measures (MMRM) with absolute change from baseline in CFQ-R respiratory domain score at each post-baseline visit as the dependent variable. The model will include treatment group, visit, and treatment-by-visit interaction as fixed effects, and will be adjusted for selected covariates as appropriate. Details will be described in the SAP. The model will be estimated using restricted maximum likelihood. Denominator degrees of freedom for the F test for fixed effects will be estimated using the Kenward-Roger approximation. An unstructured covariance structure will be used to model the within-subject errors. If the model

estimation does not converge, a compound symmetry covariance structure will be used instead. Conditional on the observed data and covariates, missing data will be assumed to be missing at random; consequently, no imputation of missing data will be performed.

The primary result obtained from the model will be the estimated treatment difference through Week 24 (defined as the average of Weeks 4, 8, 16, 24). The least squares (LS) mean estimate with a 2-sided 95% CI and a 2-sided *P* value will be provided. The treatment difference at each post-baseline visit, obtained from the model, will also be provided.

Additional or subgroup analyses if appropriate will be described in the SAP.

## 12.3.3.2 Analysis of Key Secondary Endpoint

## • Absolute change in ppFEV<sub>1</sub> from baseline through Week 24

The analysis of this endpoint will be based on an MMRM model similar to the CFQ-R endpoint above, with absolute change from baseline in ppFEV<sub>1</sub> at each post-baseline visit as the dependent variable.

The primary result obtained from the model will be the estimated treatment difference through Week 24 (defined as the average of Weeks 4, 8, 16, 24). Data obtained from the Day 15, Week 4, Week 8, Week 16, and Week 24 Visits will be included in the model. The Day 15 Visit will not be included in the estimation of the average treatment effect through Week 24. The LS mean estimate with a 2-sided 95% CI and a 2-sided *P* value will be provided. The treatment difference at each post-baseline visit, obtained from the model, will also be provided.

## 12.3.3.3 Analysis of Secondary Endpoint

## • Absolute change in SwCl from baseline through Week 24

The analysis of this endpoint will be based on an MMRM model similar to the analysis of the primary endpoints above, with absolute change from baseline in SwCl at each post-baseline visit as the dependent variable. Data obtained from Week 4, Week 8, and Week 24 Visits will be included in the model and all of these visits will be included in the estimation of the average treatment effect through Week 24. The treatment difference at each post-baseline visit, obtained from the model will also be provided.

## 12.3.3.4 Multiplicity Adjustment

A hierarchical fixed-sequence testing procedure will be used to control the overall family-wise type I error at a 2-sided alpha of 0.05 for the testing of the primary endpoint and key secondary endpoints. The testing order is as follows:

- 1. Primary endpoint: Absolute change in CFQ-R respiratory domain score from baseline through Week 24
- 2. Key secondary endpoint: Absolute change in ppFEV<sub>1</sub> from baseline through Week 24

For a test at any step to be considered statistically significant within the testing hierarchy, it must be statistically significant, and all previous tests (if any) within the hierarchy must be statistically significant. In other words, the key secondary endpoint (ppFEV<sub>1</sub>) will only be tested if the primary endpoint is statistically significant.

## 12.3.4 Safety Analysis

All safety analyses will be based on data from the TE Period for all subjects in the Safety Set.

The overall safety profile of study drug will be assessed based on the following safety and tolerability endpoints:

- Treatment-emergent adverse events (TEAEs)
- Clinical laboratory values (i.e., hematology, serum chemistry, coagulation, and urinalysis)
- ECGs
- Vital signs
- Pulse oximetry

All safety data from the TE Period will be summarized by treatment group, unless otherwise specified.

All safety data will be presented in individual subject data listings, including safety data from the Run-in Period.

### 12.3.4.1 Adverse Events

For analysis purposes, AEs will be classified as pretreatment AEs, TEAEs during the Run-in Period, TEAEs during the Treatment Period, or post-treatment AEs, defined as follows:

- **Pretreatment AE**: any AE that occurred before the first dose date of study drug (TEZ/IVA) in the Run-in Period
- **TEAE during the Run-in Period**: any AE that worsened (either in severity or seriousness) or that was newly developed at or after the first dose date of study drug (TEZ/IVA) through the end of the TE Period for the Run-in Period
- TEAE during the Treatment Period: any AE that worsened (either in severity or seriousness) or that was newly developed at or after the first dose date of study drug (TC or placebo + TEZ/IVA) in the Treatment Period through the end of the TE Period for the Treatment Period
- **Post-treatment AE**: any AE that worsened (either in severity or seriousness) or that was newly developed after:
  - o the TE Period for the Run-in Period if the subject did not receive treatment in the Treatment Period
  - o the TE Period for the Treatment Period if the subject received treatment in the Treatment Period

For AEs with missing or partial start dates, if there is no clear evidence that the AEs started before or after study drug treatment, then the AEs will be classified as TEAEs corresponding to the Treatment Period.

Unless otherwise specified, TEAE refers to TEAE during the Treatment Period.

AE summary tables will be presented by treatment group, and will include the following:

Overview of TEAEs

- TEAEs
- Related TEAEs
- TEAEs by maximum severity
- Grade 3/4 TEAEs
- Serious TEAEs
- Related serious TEAEs
- AE of special interest (details will be described in SAP)
- TEAEs leading to treatment discontinuation
- TEAEs leading to treatment interruption

Summaries will be presented by MedDRA SOC and PT using frequency counts and percentages (i.e., number and percentage of subjects with an event). When summarizing the number and percentage of subjects with an event, subjects with multiple occurrences of the same AE or a continuing AE will be counted once, only the maximum severity level will be presented in the severity summaries, and the strongest relationship level in the relationship summaries.

Listings containing individual subject level AE data will be provided separately for:

- Serious TEAEs
- TEAEs leading to treatment discontinuation
- TEAEs leading to treatment interruption
- TEAEs leading to death

In addition, all AEs, including pre- and post-treatment AEs, will be presented in individual subject data listings.

## 12.3.4.2 Clinical Laboratory Assessments

For the treatment-emergent laboratory measurements, the observed values and change from baseline values of the continuous hematology, serum chemistry, and coagulation results will be summarized in SI units by treatment group at each visit.

The number and percentage of subjects with at least 1 threshold analysis event during the TE Period will be summarized by treatment group. The threshold analysis criterion shift from baseline will also be summarized for select laboratory parameters. The threshold analysis criteria and the parameter selection criteria will be provided in the SAP.

Results of urinalysis and pregnancy tests will be listed in individual subject data listings only. In addition, a listing containing individual subject hematology, chemistry, and coagulation values will be provided. This listing will include data from scheduled and unscheduled visits.

## 12.3.4.3 Electrocardiogram

For the treatment-emergent ECG measurements, a summary of observed values and change from baseline values will be provided by treatment group, at each visit and time point, as applicable, for the following ECG interval measurements (in msec): RR, PR, QT, and QT corrected for heart rate (QTcF), QRS duration, and HR (beats per minute).

The number and percentage of subjects with at least 1 threshold analysis event during the TE Period will be summarized by treatment group. The threshold analysis criteria will be provided in the SAP.

Additional ECG analyses may be described in the SAP.

### **12.3.4.4 Vital Signs**

For the treatment-emergent vital signs measurements, the observed values and change from baseline values will be summarized by treatment group at each visit. The following vital signs parameters will be summarized: systolic and diastolic blood pressure (mm Hg), body temperature (°C), pulse rate (beats per minute), and respiratory rate (breaths per minute).

The number and percentage of subjects with at least 1 threshold analysis event during the TE Period will be summarized by treatment group. The threshold analysis criteria will be provided in the SAP.

Additional vital signs analyses may be described in the SAP.

### 12.3.4.5 Pulse Oximetry

For the treatment-emergent pulse oximetry measurements, a summary of observed values and change from baseline values will be provided by treatment group, at each visit for the percent of oxygen saturation by pulse oximetry.

The number and percentage of subjects with shift changes from baseline (normal/missing and low according to the reference range) to the lowest percent of oxygen saturation during the TE Period will be summarized by treatment group.

## 12.3.4.6 Physical Examination

PE findings will be presented in an individual subject data listing only.

### 12.3.5 Interim and IDMC Analyses

### 12.3.5.1 Interim Analysis

An IA may be performed when approximately 70% subjects complete the Week 24 Visit. To control the family-wise type 1 error rate, O'Brien-Fleming<sup>20</sup> group sequential boundaries will be applied. Specifically, if the number of subjects included in the IA is 108, the null hypotheses will be tested at a 2-sided significance level of 0.014 at the IA and 0.046 at final analysis. The actual boundaries at the IA and final analysis will be calculated based on the number of actual subjects included in the IA.

The Vertex Biometrics team will assign an internal biostatistician independent of the study team or a designated independent third-party vendor to perform the IA. The assigned independent statistician/vendor will not be involved in or influence the conduct of the study.

### 12.3.5.2 IDMC Analysis

Not applicable.

## 13 PROCEDURAL, ETHICAL, REGULATORY, AND ADMINISTRATIVE CONSIDERATIONS

# 13.1 Adverse Event and Serious Adverse Event Documentation, Severity Grading, and Reporting

### 13.1.1 Adverse Events

### 13.1.1.1 Definition of an Adverse Event

An AE is defined as any untoward medical occurrence in a subject during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or worsening of a pre-existing condition (e.g., increase in its severity or frequency) after the ICF is signed.

An AE is considered serious if it meets the definition in Section 13.1.2.1.

### 13.1.1.2 Clinically Significant Assessments

Study assessments including laboratory tests, ECGs, PEs, and vital signs will be assessed and those deemed to have clinically significant worsening from baseline will be documented as an AE. When possible, a clinical diagnosis for the study assessment will be provided, rather than the abnormal test result alone (e.g., urinary tract infection, anemia). In the absence of a diagnosis, the abnormal study assessment itself will be listed as the AE (e.g., bacteria in urine or decreased hemoglobin).

An abnormal study assessment is considered clinically significant if the subject has 1 or more of the following:

- Concomitant signs or symptoms related to the abnormal study assessment
- Further diagnostic testing or medical/surgical intervention
- A change in the dose of study drug or discontinuation from the study

Repeat testing to determine whether the result is abnormal, in the absence of any of the above criteria, does not necessarily meet clinically significant criteria. The determination of whether the study assessment results are clinically significant will be made by the investigator.

A laboratory value that is Grade 4 will not automatically be an SAE. A Grade 4 laboratory value will be an SAE if the subject's clinical status indicates a life-threatening AE.

### 13.1.1.3 Documentation of Adverse Events

All AEs will be collected from the time the ICF is signed until the subject completes study participation, as defined in Section 9.1.7

All subjects will be queried, using nonleading questions, about the occurrence of AEs at each study visit. When possible, a constellation of signs and/or symptoms will be identified as 1 overall event or diagnosis. All AEs for enrolled subjects will be recorded in the CRF and source document. AEs for subjects who are screened but not subsequently enrolled will be recorded only in the subject's source documents. The following data will be documented for each AE:

• Description of the event

- Classification of "serious" or "nonserious"
- Date of first occurrence and date of resolution (if applicable)
- Severity
- Causal relationship to study drug(s)
- Action taken
- Outcome
- Concomitant medication or other treatment given

## 13.1.1.4 Adverse Event Severity

The investigator will determine and record the severity of all serious and nonserious AEs. The guidance available at the following website will be consulted: Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0, Cancer Therapy Evaluation Program, http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm (Accessed February 2019). AEs of CTCAE Grades 4 and 5 will be documented as "life-threatening." When considering the severity of an AE in a pediatric subject, the investigator will consider that reference ranges for pediatric clinical laboratory parameters may differ from those in the CTCAE. The severity of an AE described by a term that does not appear in the CTCAE will be determined according to the definitions in Table 13-1.

**Table 13-1** Grading of AE Severity

| Classification | Definition |
|---|---|
| Mild (Grade 1) | Mild level of discomfort and does not interfere with regular activities |
| Moderate (Grade 2) Moderate level of discomfort and significantly interferes with regula | |
| Severe (Grade 3) | Significant level of discomfort and prevents regular activities |
| Life-threatening (Grade 4) | Any adverse drug event that places the subject, in the view of the investigator, at immediate risk of death |

AE: adverse event

## 13.1.1.5 Adverse Event Causality

Every effort will be made by the investigator to assess the relationship of the AE, if any, to the study drug(s). Causality will be classified using the categories in Table 13-2.

Table 13-2 Classifications for AE Causality

| Classification | Definition |
|---|---|
| Related | There is an association between the event and the administration of investigational study drug, a plausible mechanism for the event to be related to the investigational study drug and causes other than the investigational study drug have been ruled out, and/or the event reappeared on re-exposure to the investigational study drug. |
| Possibly related | There is an association between the event and the administration of the investigational study drug and there is a plausible mechanism for the event to be related to investigational study drug, but there may also be alternative etiology, such as characteristics of the subject's clinical status or underlying disease. |
| Unlikely related | The event is unlikely to be related to the investigational study drug and likely to be related to factors other than investigational study drug. |

Table 13-2 Classifications for AE Causality

| Classification | Definition |
|---|---|
| Not related | The event is related to an etiology other than the investigational study drug (the |
| | alternative etiology will be documented in the subject's medical record). |

AE: adverse event

## 13.1.1.6 Study Drug Action Taken

The investigator will classify the study drug action taken with regard to the AE. The action taken will be classified according to the categories in Table 13-3.

Table 13-3 Classifications for Study Drug Action Taken With Regard to an AE

| Classification | Definition Study drug dose not changed in response to an AE |
|---|---|
| Dose not changed | |
| Dose reduced | Study drug dose reduced in response to an AE |
| <b>Drug interrupted</b> Study drug administration interrupted in response to an AE | |
| Drug withdrawn | Study drug administration permanently discontinued in response to an AE |
| Not applicable | Action taken regarding study drug administration does not apply. |
| | "Not applicable" will be used in circumstances such as when the investigational treatment had been completed before the AE began and no opportunity to decide whether to continue, interrupt, or withdraw treatment is possible. |

AE: adverse event

### 13.1.1.7 Adverse Event Outcome

An AE will be followed until the investigator has determined and provided the final outcome. The outcome will be classified according to the categories in Table 13-4.

Table 13-4 Classifications for Outcome of an AE

| Classification | Definition |
|---|---|
| Recovered/resolved | Resolution of an AE with no residual signs or symptoms |
| Recovered/resolved with sequelae | Resolution of an AE with residual signs or symptoms |
| Not recovered/not resolved (continuing) | Either incomplete improvement or no improvement of an AE, such that it remains ongoing |
| Fatal | Outcome of an AE is death. "Fatal" will be used when death is at least possibly related to the AE. |
| Unknown | Outcome of an AE is not known (e.g., a subject lost to follow up) |

AE: adverse event

### 13.1.1.8 Treatment Given

The investigator ensures adequate medical care is provided to subjects for any AEs, including clinically significant laboratory values related to study drug. In addition, the investigator will describe whether any treatment was given for the AE. "Yes" is used if any treatment was given in response to an AE, and may include treatments such as other medications, surgery, or physical therapy. "No" indicates the absence of any kind of treatment for an AE.

### 13.1.2 Serious Adverse Events

### 13.1.2.1 Definition of a Serious Adverse Event

An SAE is any AE that meets any of the following outcomes:

- Fatal (death, regardless of cause, that occurs during participation in the study or occurs after participation and is suspected of being a delayed toxicity due to administration of the study drug)
- Life-threatening, such that the subject was at immediate risk of death from the reaction as it occurred
- Inpatient hospitalization or prolongation of hospitalization
- Persistent or significant disability/incapacity (disability is defined as a substantial disruption of a person's ability to conduct normal life functions)
- Congenital anomaly or birth defect
- Important medical event that, based upon appropriate medical judgment, may jeopardize the subject or may require medical or surgical intervention to prevent 1 of the outcomes listed above (e.g., an allergic bronchospasm requiring intensive treatment in an emergency room or at home)

If a subject has a hospitalization or procedure (e.g., surgery) for an event or condition that occurred before the subject signed the ICF, and the hospitalization or procedure was planned before the subject signed the ICF, the hospitalization or procedure will not be considered to indicate an SAE, unless an AE caused the hospitalization or procedure to be rescheduled sooner or to be prolonged relative to what was planned. In addition, hospitalizations clearly not associated with an AE (e.g., social hospitalization for purposes of respite care) will not be considered to indicate an SAE.

Clarification will be made between the terms "serious" and "severe" because they are not synonymous. The term "severe" is often used to describe the intensity (severity) of a specific event, as in mild, moderate, or severe myocardial infarction. The event itself, however, may be of relatively minor medical significance, such as a severe headache. This is not the same as "serious", which is based on subject/event outcome or action described above, and is usually associated with events that pose a threat to a subject's life or functioning. Seriousness, not severity, serves as a guide for defining expedited regulatory reporting obligations.

## 13.1.2.2 Reporting and Documentation of Serious Adverse Events

All SAEs that occur after obtaining informed consent and assent (where applicable) through the completion of study participation, regardless of causality, will be reported by the investigator to Vertex GPS within 24 hours of identification. In addition, all SAEs that occur after the completion of study participation and are considered related to study drug(s) will be reported to Vertex GPS within 24 hours of identification.

For SAEs that occur after obtaining informed consent and assent (where applicable) through the completion of study participation, the SAE Form will be completed for new/initial events as well as to report follow-up information on previously reported events. Investigators are asked to report follow-up information as soon as it becomes available to ensure timely reporting to health authorities.

| Please send completed SAE Forms to | Vertex GPS via: |
|------------------------------------|--------------------|
| Email: | (preferred choice) |
| Fax: | |

For technical issues related to submitting the form, contact telephone:

SAEs that occur after the completion of study participation and are considered related to study drug(s) will be recorded on the Vertex Clinical Trial Safety Information Collection Form (hereafter referred to as the "SAE Form") using a recognized medical term or diagnosis that accurately reflects the event. SAEs will be assessed by the investigator for relationship to the investigational study drug(s) and possible etiologies. On the SAE Form, relationship to study drug(s) will be assessed only as related (includes possibly related) or not related (includes unlikely related), and severity assessment will not be required. For the purposes of study analysis, if the event has not resolved at the end of the study reporting period, it will be documented as ongoing. For purposes of regulatory safety monitoring, the investigator is required to follow the event to resolution and report the outcome to Vertex using the SAE Form.

## 13.1.2.3 Expedited Reporting and Investigator Safety Letters

Vertex, as study sponsor, is responsible for reporting suspected, unexpected, serious adverse reactions (SUSARs) involving the study drug(s) to all regulatory authorities, IECs, and participating investigators in accordance with ICH Guidelines and/or local regulatory requirements, as applicable. In addition, Vertex, or authorized designee, will be responsible for the submission of safety letters to central IECs.

It is the responsibility of the investigator or designee to promptly notify the local IRB/ IEC of all unexpected serious adverse drug reactions involving risk to human subjects.

## 13.2 Administrative Requirements

### 13.2.1 Ethical Considerations

The study will be conducted in accordance with the current ICH GCP Guidelines, which are consistent with the ethical principles founded in the Declaration of Helsinki, and in accordance with local applicable laws and regulations. The IRB/IEC will review all appropriate study documentation to safeguard the rights, safety, and well-being of the subjects. The study will be conducted only at sites where IRB/IEC approval has been obtained. The protocol, Investigator's Brochure, sample ICF, advertisements (if applicable), written information given to the subjects (including diary cards), safety updates, annual progress reports, and any revisions to these documents will be provided to the IRB/IEC by the investigator or Vertex, as allowable by local applicable laws and regulations.

## 13.2.2 Subject Information and Informed Consent

After the study has been fully explained, written informed consent will be obtained from the subject or legal representative or guardian (if applicable), and assent will be obtained from the subject (if applicable), before study participation. The method of obtaining and documenting the informed consent and assent (if applicable) and the contents of the consent will comply with ICH GCP and all applicable laws and regulations and will be subject to approval by Vertex or its designee.

## 13.2.3 Investigator Compliance

No modifications to the protocol will be made without the approval of both the investigator and Vertex. Changes that significantly affect the safety of the subjects, the scope of the investigation, or the scientific quality of the study (i.e., efficacy assessments) will require IRB/IEC notification before implementation, except where the modification is necessary to eliminate an apparent immediate hazard to human subjects. Vertex will submit all protocol modifications to the required regulatory authorities.

When circumstances require an immediate departure from procedures set forth in the protocol, the investigator will contact Vertex to discuss the planned course of action. If possible, contact will be made before the implementation of any changes. Any departures from the protocol will be fully documented in the source documentation and in a protocol deviation log.

### 13.2.4 Access to Records

The investigator will make the office and/or hospital records of subjects enrolled in this study available for inspection by Vertex or its representative at the time of each monitoring visit and for audits. The records will also be available for direct inspection, verification, and copying, as required by applicable laws and regulations, by officials of the regulatory health authorities (FDA and others). The investigator will comply with applicable privacy and security laws for use and disclosure of information related to the research set forth in this protocol.

## 13.2.5 Subject Privacy

To maintain subject confidentiality and to comply with applicable data protection and privacy laws and regulations, all data provided to Vertex, study reports, and communications relating to the study will identify subjects by assigned subject numbers, and access to subject names linked to such numbers will be limited to the site and the study physician and will not be disclosed to Vertex. As required by applicable laws and regulations in the countries in which the study is being conducted, the investigator will allow Vertex and/or its representatives access to all pertinent medical records to allow for the verification of data gathered and the review of the data collection process. The FDA and regulatory authorities in other jurisdictions, including the IRB/IEC, may also request access to all study records, including source documentation, for inspection.

### 13.2.6 Record Retention

The investigator will maintain all study records according to ICH GCP Guidelines and/or applicable local regulatory requirement(s), whichever is longest, as described in the Clinical Trial Agreement. If the investigator withdraws from the responsibility of keeping the study records, custody will be transferred to a person willing to accept the responsibility and Vertex will be notified.

### 13.2.7 Study Termination

At any time, Vertex may terminate this study in its entirety or may terminate this study at any particular site. In addition, for reasonable cause, either the investigators or their IRBs/IECs may terminate the study at their center.

Conditions that may lead to reasonable cause and warrant termination include, but are not limited to:

- Subject or investigator noncompliance
- Unsatisfactory subject enrollment
- Lack of adherence to protocol procedures
- Lack of evaluable and/or complete data
- Potentially unacceptable risk to study subjects
- Decision to modify drug development plan
- Decision by the FDA or other regulatory authority

Written notification that includes the reason for the clinical study termination is required.

## 13.2.8 End of Study

The end of study is defined as the last scheduled visit (or scheduled contact) of the last subject.

### 13.3 Data Quality Assurance

Vertex or its designated representative will conduct a study site visit to verify the qualifications of each investigator, inspect clinical study site facilities, and inform the investigator of responsibilities and procedures for ensuring adequate and correct study documentation. Vertex will provide, or assess and approve, any electronic data capture (EDC) tools.

The investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the study for each subject. Data collected during the study, including results from screening, will be recorded in a data capture system for each enrolled subject. Each subject's set of captured data records, once complete, will be signed and dated by the investigator.

### 13.4 Monitoring

Monitoring and auditing procedures developed or approved by Vertex will be followed to comply with GCP Guidelines. On-site checking of the data captured for the study/SAE Forms for completeness and clarity, and clarification of administrative matters will be performed.

The study will be monitored by Vertex or its designee. Monitoring will be done by personal visits from a representative of Vertex or designee (study site monitor), who will review the data captured for the study/SAE Forms and source documents. The study site monitor will ensure that the investigation is conducted according to the protocol design and regulatory requirements.

## 13.5 Electronic Data Capture

Sites will use an EDC tool to record data for each enrolled subject.

It is the investigator's responsibility to ensure the accuracy, completeness, clarity, and timeliness of the data reported. The investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the study for each subject, including the dates and details of study procedures, AEs, other observations, and subject status.

The audit trail entry will show the user's identification information and the date and time of any correction. The investigator will provide formal approval of all data reported to Vertex, including

any changes made, to endorse the final submitted data for the subjects for whom the investigator is responsible.

## 13.6 Confidentiality and Disclosure

Any and all scientific, commercial, and technical information disclosed by Vertex in this protocol or elsewhere will be considered the confidential and proprietary property of Vertex. The investigator shall hold such information in confidence and shall not disclose the information to any third party except to such of the investigator's employees and staff as have been made aware that the information is confidential and who are bound to treat it as such and to whom disclosure is necessary to evaluate that information. The investigator shall not use such information for any purpose other than determining mutual interest in performing the study and, if the parties decide to proceed with the study, for the purpose of conducting the study.

The investigator understands that the information developed from this clinical study will be used by Vertex in connection with the development of the study drug and other drugs and diagnostics, and therefore may be disclosed as required to other clinical investigators, business partners and associates, the FDA, and other government agencies. The investigator also understands that, to allow for the use of the information derived from the clinical study, the investigator has the obligation to provide Vertex with complete test results and all data developed in the study.

## 13.7 Publications and Clinical Study Report

## 13.7.1 Publication of Study Results

Vertex is committed to reporting the design and results of all clinical studies in a complete, accurate, balanced, transparent, and timely manner, consistent with Good Publication Practices (GPP3).<sup>21</sup>

**Publication Planning**: Vertex staff along with the lead principal investigators, the steering committee, and/or the publication committee will work together to develop a publication plan.

**Authorship**: Authorship of publications will be determined based on the Recommendations for Conduct, Reporting, Editing, and Publication of Scholarly Work in Medical Journals, which states that authorship should be based on the following 4 criteria<sup>22</sup>:

- 1. Substantial contributions to conception and design, acquisition of data, or analysis and interpretation of data;
- 2. Drafting of the article or revising it critically for important intellectual content;
- 3. Final approval of the version to be published; and
- 4. Agreement to be accountable for all aspects of the work in ensuring that questions related to the accuracy or integrity of any part of the work are appropriately investigated and resolved.

All authors must meet conditions 1, 2, 3, and 4. All persons designated as authors should qualify for authorship, and all those who qualify should be listed. Contributions such as medical writing, enrollment of subjects, acquisition of funding, collection of data, or general supervision of the research group, alone, do not justify authorship.

**Contributors**: Contributors who meet fewer than all 4 of International Committee of Medical Journal Editors (ICMJE) criteria for authorship will not be listed as authors, but their

contribution will be acknowledged and specified either as a group (e.g., "study investigators") or individually (e.g., "served as scientific advisor").

**Publication Review**: As required by a separate clinical study agreement, Vertex must have the opportunity to review all publications, including any manuscripts, abstracts, oral/slide presentations, and book chapters regarding this study before submission to congresses or journals for consideration.

## 13.7.2 Clinical Study Report

A CSR, written in accordance with the ICH E3 Guideline, will be submitted in accordance with local regulations.

### 14 REFERENCES

- 1 Cystic Fibrosis Foundation. What is cystic fibrosis? Available at: https://www.cff.org/What-is-CF/About-Cystic-Fibrosis/. Accessed 22 March 2018.
- 2 Cystic Fibrosis Foundation. Patient Registry: 2017 Annual Data Report. Bethesda, MD: Cystic Fibrosis Foundation; 2018.
- 3 European Cystic Fibrosis Society. 2016 ECFS Patient Registry Annual Data Report. Karup, Denmark: European Cystic Fibrosis Society; 2018.
- 4 United States Department of Health and Human Services. Food and Drug Administration. Office of Orphan Products Development. Developing Products for Rare Diseases & Conditions. Available at: http://www.fda.gov/ForIndustry/DevelopingProductsforRareDiseasesConditions/default. htm. Accessed 19 September 2016.
- 5 European Medicines Agency [Internet]. Committee for Orphan Medicinal Products (COMP). Available at: https://www.ema.europa.eu/en/committees/committee-orphan-medicinal-products-comp. Accessed 07 December 2018.
- Rommens J, Iannuzzi M, Kerem B, Drumm M, Melmer G, Dean M, et al. Identification of the cystic fibrosis gene: chromosome walking and jumping. Science. 1989;245(4922):1059-65.
- 7 Kreindler JL. Cystic fibrosis: exploiting its genetic basis in the hunt for new therapies. Pharmacol Ther. 2010;125(2):219-29.
- 8 Sheppard MN, Nicholson AG. The pathology of cystic fibrosis. Curr Diagn Pathol. 2002;8(1):50-59.
- 9 Flume PA, VanDevanter DR. State of progress in treating cystic fibrosis respiratory disease. BMC Med. 2012;10(1):88.
- 10 CFTR2.org. Clinical and functional translation of CFTR. The Clinical and Functional TRanslation of CFTR (CFTR2), US Cystic Fibrosis Foundation, Johns Hopkins University, the Hospital for Sick Children. Available at: http://www.cftr2.org. Accessed 09 January 2018.
- Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, et al. Multi-ethnic reference values for spirometry for the 3–95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012;40(6):1324-43.
- Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, et al. Standardisation of spirometry. Eur Respir J. 2005;26(2):319-38.
- Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation.

  Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999;130(6):461-70
- Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, et al. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006;145(4):247-54.
- 15 Counahan R, Chantler C, Ghazali S, Kirkwood B, Rose F, Barratt TM. Estimation of glomerular filtration rate from plasma creatinine concentration in children. Arch Dis Child. 1976;51(11):875-78.

- Goss CH, Quittner AL. Patient-reported outcomes in cystic fibrosis. Proc Am Thorac Soc. 2007;4(4):378-86.
- Quittner AL, Buu A, Messer MA, Modi AC, Watrous M. Development and validation of the Cystic Fibrosis Questionnaire in the United States. Chest. 2005;128(4):2347-54.
- Henry B, Aussage P, Grosskopf C, Goehrs JM. Development of the Cystic Fibrosis Questionnaire (CFQ) for assessing quality of life in pediatric and adult patients. Qual Life Res. 2003;12(1):63-76.
- Wenninger K, Aussage P, Wahn U, Staab D, German Cystic Fibrosis Questionnaire study group. The revised German Cystic Fibrosis Questionnaire: validation of a disease-specific health-related quality of life instrument. Qual Life Res. 2003;12(1):77-85.
- O'Brien PC, Fleming TR. A Multiple Testing Procedure for Clinical Trials. Biometrics. 1979;35(3):549-56.
- Battisti WP, Wager E, Baltzer L, Bridges D, Cairns A, Carswell CI, et al. Good Publication Practice for Communicating Company-Sponsored Medical Research: GPP3. Ann Intern Med. 2015;163(6):461-4.
- 22 (ICMJE). ICoMJE. Recommendations for conduct, reporting, editing, and publication of scholarly work in medical journals. [Internet]. Available from: Accessed April 9,.

## 15 PROTOCOL SIGNATURE PAGES

## 15.1 Sponsor Signature Page

| Protocol #: | VX18-445-109 | Version #: | 1.0 | Version Date: | 30 May 2019 |
|---|---|---|---|---|---|
| Study Title: A Phase 3b, Randomized, Double-blind, Controlled Study Evaluating the Efficacy | | | | | |
| and Safety of VX-445/Tezacaftor/Ivacaftor in Cystic Fibrosis Subjects, Homozygous for | | | | | |
| F508del | | | | | |

This Clinical Study Protocol has been reviewed and approved by the sponsor.

## 15.2 Investigator Signature Page

| Protocol #: | VX18-445-109 | Version #: | 1.0 | Version Date: | 30 May 2019 |
|---|---|---|---|---|---|
| Study Title: A Phase 3b, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-445/Tezacaftor/Ivacaftor in Cystic Fibrosis Subjects, Homozygous for <i>F508del</i> | | | | | |
| I have read Protocol VX18-445-109, Version 1.0, and agree to conduct the study according to its terms. I understand that all information concerning VX-445, tezacaftor, and ivacaftor and this protocol supplied to me by Vertex Pharmaceuticals Incorporated (Vertex) is confidential. | | | | | |
| Printed Name | | | _ | | |
| Signature | _ | | Date | e | |